

## **Clinical Trial Protocol**

| | Document Number: | c32737758-02 |
|---|---|---|
| EudraCT No. | 2020-004388-22 | |
| BI Trial No. | 1425-0010 | |
| BI Investigational<br>Medicinal Product | BI 706321 | |
| Title | Effect of itraconazole on the pharmac dose of BI 706321 in healthy male su period fixed sequence design study) | <u>e</u> |
| Lay Title | A study in healthy men to test how its amount of BI 706321 in the blood | raconazole influences the |
| Clinical Phase | I | |
| Clinical Trial Leader | Phone:<br>Fax: | |
| Principal<br>Investigator | Phone:<br>Fax: | |
| Status | Final Protocol (Revised Protocol (bas | ed on global amendment 1)) |
| Version and Date | Version: 2.0 | Date: 01 February 2021 |
| Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies. All rights reserved. This document may not - in full or in part - be passed on, reproduced, published or otherwise used without prior written permission | | |


Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## CLINICAL TRIAL PROTOCOL SYNOPSIS

| Company name | Boehringer Ingelheim |
|---|---|
| Protocol date | 02 November 2020 |
| Revision date | 01 February 2021 |
| BI trial number | 1425-0010 |
| Title of trial | Effect of itraconazole on the pharmacokinetics of a single oral dose of BI 706321 in healthy male subjects (an open-label, two-period fixed sequence design study) |
| Principal Investigator: | |
| Trial site | |
| Clinical phase | I |
| Trial rationale | Based on <i>in vitro</i> data, CYP3A4 and P-gp are involved in metabolism and transport of BI 706321, respectively. It is therefore necessary to explore the relative bioavailability of BI 706321 in plasma when given alone versus when given together with a strong CYP3A4 and P-gp inhibitor. |
| Trial objective | To investigate the pharmacokinetics of a single oral dose of BI 706321 when given alone (treatment R) or in combination with itraconazole (treatment T) |
| Trial design | Open-label, two-treatment, two-period fixed sequence design |
| Trial endpoints: | Primary endpoints: AUC <sub>0-∞</sub> and C <sub>max</sub> of BI 706321 in plasma Secondary endpoints: AUC <sub>0-tz</sub> of BI 706321 in plasma |
| Number of subjects | |
| total entered | 14 |
| each treatment | 14 |
| Diagnosis | Not applicable |
| Main criteria<br>for inclusion | Healthy male subjects, age of 18 to 50 years (inclusive), body mass index (BMI) of 18.5 to 29.9 kg/m² (inclusive) |
| Test product 1 | BI 706321 tablet formulation tablet strength) |
| dose | as single dose |
| mode of admin. | Oral with 240 mL of water after an overnight fast of at least 10 h |

c32737758-02 Trial Protocol 

| Proprietary confidential information © 202 | Boehringer Ingelheim International GmbH | or one or more of its affiliated companies |
|---|---|---|

| Test product 2 | Itraconazole oral solution (Sempera® Liquid 10 mg/mL) |
|---|---|
| _ | |
| dose | 200 mg once daily (q.d.) |
| mode of admin. | Oral with 240 mL of water after an overnight fast of at least 9 h |
| Duration of treatment | Treatment R (BI 706321 alone): |
| | Single dose of BI 706321 (Day 1) |
| | Treatment T (itraconazole + BI 706321): |
| | 14 days of itraconazole treatment (200 mg itraconazole once daily from Day -3 to Day 11) combined with a single dose of BI 706321 on the fourth day of the itraconazole treatment (Day 1, 1 h after the itraconazole administration) |
| | Wash-out period: |
| | Administrations of BI 706321 will be separated by a wash-out phase of at least 14 days. |
| Statistical methods | Extent of drug-drug-interaction will be estimated by the ratios of the geometric means (test/reference) for the primary and secondary endpoints. Additionally, their two-sided 90% confidence intervals (CIs) will be provided. This method corresponds to the two one-sided t-test procedure, each at a 5% significance level. Since the main focus is on estimation and not testing, a formal hypothesis test and associated acceptance range are not specified. The statistical model will be an analysis of variance (ANOVA) on the logarithmic scale including effects for 'subject' and 'treatment'. CIs will be calculated based on the residual error from the ANOVA. |
| | Descriptive statistics will be calculated for all endpoints. |

c32737758-02 Trial Protocol 

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### **FLOW CHART**

| Period | Visit | Day | Planned time (relative to drug administration) | Approximate clock time of actual day [h:min] | Event and comment | Safety laboratory <sup>5</sup> | PK blood, BI 706321 | 12-lead ECG | Vital signs (Body<br>temperature, BP, PR) | Questioning for AEs and concomitant therapy 7 |
|---|---|---|---|---|---|---|---|---|---|---|
| SCR | 1 | -21 to -3 | | | Screening (SCR) <sup>1</sup> | $\mathbf{x}^{\mathbf{A}}$ | | X | X | |
| | 2 | -3 to -1 | -73:00 | 08:00 | Ambulatory visit | xB | | | | X |
| | | 1 | -3:00 | 06:00 | Admission to trial site <sup>2</sup> | $x^{2,3}$ | $\mathbf{x}^2$ | $\mathbf{x}^2$ | $\mathbf{x}^2$ | $\mathbf{x}^2$ |
| | | | 0:00 | 09:00 | BI 706321 administration | | | | | |
| | | | 0:30 | 09:30 | | | X | | | |
| | | | 1:00 | 10:00 | | | X | | | |
| )e) | | | 2:00 | 11:00 | 240 mL fluid intake | | X | | | |
| lor | | | 3:00 | 12:00 | | | X | | | |
| Period 1/ Treatment R (BI 706321 alone) <sup>8</sup> | | | 4:00 | 13:00 | 240 mL fluid intake, thereafter lunch <sup>4</sup> | | X | X | X | X |
| 632 | | | 5:00 | 14:00 | | | X | | | |
| 70 | | | 6:00 | 15:00 | | | X | | | |
| BI | | | 7:00 | 16:00 | Snack (voluntary) <sup>4</sup> | | X | | | |
| R ( | | | 8:00 | 17:00 | | | X | | | |
| int | | | 10:00 | 19:00 | Dinner <sup>4</sup> | | X | | | |
| me | | | 12:00 | 21:00 | | | X | | | X |
| eat | | 2 | 24:00 | 09:00 | Breakfast (voluntary) <sup>4</sup> , | xB | X | X | X | X |
| , T <sub>1</sub> | | | | | discharge from trial site | | | | | |
| 1 1/ | | | 34:00 | 19:00 | Ambulatory visit | | X | | | X |
| ioc | | 3 | 46:00 | 07:00 | Ambulatory visit | | X | | | X |
| Per | | 4 | 70:00 | 07:00 | Ambulatory visit | | X | | | X |
| | | 5 | 94:00 | 07:00 | Ambulatory visit | | X | | | X |
| | | 6 | 118:00 | 07:00 | Ambulatory visit | | X | | | X |
| | | 7 | 142:00 | 07:00 | Ambulatory visit | xB | X | | | X |
| | | 8 | 166:00 | 07:00 | Ambulatory visit | | X | | | X |
| | | 9 | 190:00 | 07:00 | Ambulatory visit | | X | | | X |

- Subject must be informed and written informed consent obtained prior to starting any screening procedures. Screening
  procedures include physical examination, check of vital signs, ECG, safety laboratory (including drug screening),
  demographics (including determination of body height and weight, smoking status and alcohol history), relevant
  medical history, concomitant therapy and review of inclusion/exclusion criteria.
- 2. The time is approximate; the procedure is to be performed and completed within the 3 h prior to drug administration.
- 3. Urine drug screening and alcohol breath test
- 4. If several actions are indicated at the same time, the intake of meals will be the last action.
- 5. Letters A, B, C, and D define different sets of safety laboratory examinations (for details refer to Table 5.2.3: 1)
- 6. At the end of trial visit the EoTrial examination includes physical examination, vital signs, ECG, safety laboratory, recording of AEs and concomitant therapies.
- AEs and concomitant therapies will be recorded throughout the trial, but will be specifically asked for at the times indicated in the Flow Chart above.
- 8. Administration of BI 706321 in treatment R and T will be separated by at least 14 days.
- 9. Blood collection takes place at the indicated times. Itraconazole will be administered immediately thereafter.

c32737758-02 **Trial Protocol ** 

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### FLOW CHART (cont'd)

| Period | Visit | Day | Planned time (relative to<br>drug administration)<br>[h:min] | | Event and comment | Safety laboratory <sup>5</sup> | PK blood, BI 706321 | | 12-lead ECG | Vital signs (body temperature BP, PR) | Questioning for AEs and concomitant therapy 7 |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | 3 | -3 | -73:00 | 08:00 | Ambulatory visit, itraconazole administration | x <sup>B,2,3</sup> | | | | | $\frac{x^2}{x^2}$ |
| | | -2 | -49:00 | 08:00 | Ambulatory visit, itraconazole administration | 6.2 | | | | | x <sup>2</sup> |
| | | -1 | -25:00 | 08:00 | Ambulatory visit, itraconazole administration | x <sup>C,2</sup> | | - | _ | 2 | x <sup>2</sup> |
| | | 1 | -3:00 | 06:00 | Admission to trial site <sup>2</sup> | | - | | x <sup>2</sup> | $\mathbf{x}^2$ | x <sup>2</sup> |
| | | | -1:00 | 08:00 | Itraconazole administration | | x <sup>2</sup> | - | | | |
| | | | 0:00 | 09:00 | BI 706321 administration | | | - | | | |
| | | | 0:30 | 09:30 | | | X | - | | | |
| | | | 1:00 | 10:00 | 240 1 0 :1: 4 1 | | X | - | | | |
| | | | 2:00 | 11:00 | 240 mL fluid intake | | X | - | | | |
| | | | 3:00 | 12:00 | 240 1 0 11 41 6 1 14 | | X | - | | | |
| ∞ | | | 4:00 | 13:00 | 240 mL fluid intake, thereafter lunch <sup>4</sup> | | X | - | X | X | X |
| ole) | | | 5:00 | 14:00 | | | X | - | | | |
| azc | | | 6:00 | 15:00 | C 1 ( 1 , ) <sup>4</sup> | | X | - | | | |
| con | | | 7:00<br>8:00 | 16:00<br>17:00 | Snack (voluntary) <sup>4</sup> | | X | - | | - | |
| trac | | | 10:00 | 19:00 | Dinner <sup>4</sup> | | X | - | | - | |
| + | | | 12:00 | 21:00 | Dinner | | X | - | | | |
| 21 | | 2 | 23:00 | 08:00 | Itraconazole administration | | X | - | | | x<br>x <sup>2</sup> |
| 963 | | 2 | 24:00 | 09:00 | Breakfast <sup>4</sup> | | х | - | | | X |
| 1 7 | | | 28:00 | 13:00 | Lunch <sup>4</sup> | | Λ | - | | | X |
| (B | | | 31:00 | 16:00 | Snack (voluntary) <sup>4</sup> | | | - | | | Λ |
| t T | | | 34:00 | 19:00 | Dinner <sup>4</sup> | | Х | - | | | X |
| Jen | | 3 | 46:00 | 07:00 | Itraconazole administration, | x <sup>B,2</sup> | x <sup>9</sup> | - | x <sup>2</sup> | $\mathbf{x}^2$ | $\mathbf{x}^2$ |
| Period 2/ Treatment T (BI 706321 $+$ itraconazole) $^8$ | | 3 | | | discharge from trial site | Α | | | Λ | Λ | |
| , T <sub>1</sub> | | 4 | 70:00 | 07:00 | Ambulatory visit, itraconazole administration | | x <sup>9</sup> | | | | $\mathbf{x}^2$ |
| 12/ | | 5 | 94:00 | 07:00 | Ambulatory visit, itraconazole administration | x <sup>C,2</sup> | x <sup>9</sup><br>x <sup>9</sup><br>x <sup>9</sup> | | | | $ \begin{array}{c} x^2 \\ x^2 \\ x^2 \\ x^2 \\ x^2 \\ x^2 \\ x^2 \end{array} $ |
| ij | | 6 | 118:00 | 07:00 | Ambulatory visit, itraconazole administration | | x <sup>9</sup> | | | | $\mathbf{x}^2$ |
| Pe | | 7 | 142:00 | 07:00 | Ambulatory visit, itraconazole administration | x <sup>B,2</sup> | x <sup>9</sup> | | | | $\mathbf{x}^2$ |
| | | 8 | 166:00 | 07:00 | Ambulatory visit, itraconazole administration | | x <sup>9</sup> | | | | x <sup>2</sup> |
| | | 9 | 190:00 | 07:00 | Ambulatory visit, itraconazole administration | | x <sup>9</sup> | | | | <b>x</b> <sup>2</sup> |
| | | 10 | 214:00 | 07:00 | Ambulatory visit, itraconazole administration | x <sup>C,2</sup> | x <sup>9</sup> | | | | |
| | | 11 | 238:00 | 07:00 | , , | | | | | | x <sup>2</sup> |
| | | 12 | 262:00 | 07:00 | Ambulatory visit | | X | | | | X |
| | | 14 | 310:00 | 07:00 | Ambulatory visit | x <sup>C</sup> | X | | | | X |
| | | 16 | 358:00 | 07:00 | Ambulatory visit | | X | | | | X |
| | | 18 | 406:00 | 07:00 | Ambulatory visit | | X | | | | X |
| | | 20 | 454:00 | 07:00 | Ambulatory visit | | X | | | | X |
| | | 22 | 502:00 | 07:00 | Ambulatory visit | | X | | | | X |
| | | 24 | 550:00 | 07:00 | Ambulatory visit | ъ. | X | | | | X |
| FU | 4 | 25 to 35 | | | End of trial (EoTrial) examination <sup>6</sup> | $\mathbf{x}^{\mathrm{D}}$ | | | X | X | X |

- 1. Subject must be informed and written informed consent obtained prior to starting any screening procedures. Screening procedures include physical examination, check of vital signs, ECG, safety laboratory (including drug screening), demographics (including determination of body height and weight, smoking status and alcohol history), relevant medical history, concomitant therapy and review of inclusion/exclusion criteria.
- 2. The time is approximate; the procedure is to be performed and completed within the 3 h prior to drug administration.3. Urine drug screening and alcohol breath test
- 4. If several actions are indicated at the same time, the intake of meals will be the last action.

Boehringer Ingelheim BI Trial No.: 1425-0010

c32737758-02

01 Feb 2021


Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

- 5. Letters A, B, C, and D define different sets of safety laboratory examinations (for details refer to Table 5.2.3: 1)
- 6. At the end of trial visit the EoTrial examination includes physical examination, vital signs, ECG, safety laboratory, recording of AEs and concomitant therapies.
- 7. AEs and concomitant therapies will be recorded throughout the trial, but will be specifically asked for at the times indicated in the Flow Chart above.
- 8. Administration of BI 706321 in treatment R and T will be separated by at least 14 days.

**Trial Protocol** 

9. Blood collection takes place at the indicated times. Itraconazole will be administered immediately thereafter.

c32737758-02 Trial Protocol


Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## **TABLE OF CONTENTS**

| TIT | LE P | PAGE | ••••• | | 1 |
|---|---|---|---|---|---|
| CL | INIC | AL TR | IAL PR | OTOCOL SYNOPSIS | 2 |
| FLO | ) WC | CHART | Γ | | 4 |
| | | | | [S | |
| 1. | | | | | |
| | 1.1 | | | CKGROUND | |
| | 1.2 | | | <u></u> | |
| | | 1.2.1 | | 21 | |
| | | 1.2.2 | | azolel Effect Period | |
| | 1.2 | 1.2.3 | | | |
| | 1.3 | | | FOR PERFORMING THE TRIAL | |
| | 1.4 | | | SK ASSESSMENTre-related risks | |
| | | 1.4.1<br>1.4.2 | | elated risks and safety measures | |
| | | 1,4,4 | 1.4.2.1 | | |
| | | | | BI 706321 | |
| | | | 1.1.2.2 | 1.4.2.2.1 Drug-related events observed in clinical trials with | |
| | | | | 706321 | |
| | | | | 1.4.2.2.2 Risk assessment in the context of SARS-CoV-2 | |
| | | | | infection | |
| | | | | 1.4.2.2.3 Events predicted based on pharmacological proper | |
| | | | 1 4 2 2 | / preclinical information | |
| | | | 1.4.2.3 | Itraconazole | 19 |
| | | | 1.4.2.4 | Potential drug-drug interaction between BI 706321 and itraconazole | 19 |
| 2. | TDI | AI OB | e IFCTI | VES AND ENDPOINTS | |
| 4. | 2.1 | | | ΓIVES, PRIMARY AND SECONDARY ENDPOINTS | |
| | 2.1 | 2.1.1 | | ojectivesojectives | |
| | | 2.1.2 | | y endpoints | |
| | | 2.1.3 | - | ary endpoint | |
| | | | 2.2.2.2 | Safety and tolerability | |
| 3. | DES | CRIP | TION O | F DESIGN AND TRIAL POPULATION | . 23 |
| | 3.1 | OVER | ALL TR | IAL DESIGN AND PLAN | 23 |

c32737758-02 Trial Protocol

**** 

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| | 3.2 | | USSION OF TRIAL DESIGN, INCLUDING THE CHOICE OF TROL GROUPS | 23 |
|---|---|---|---|---|
| | 3.3 | | CTION OF TRIAL POPULATION | |
| | 0.0 | 3.3.1 | Main diagnosis for trial entry | |
| | | 3.3.2 | Inclusion criteria | |
| | | 3.3.3 | Exclusion criteria | |
| | | | Withdrawal of subjects from treatment or assessments | |
| | | | 3.3.4.1 Discontinuation of trial treatment | |
| | | | 3.3.4.2 Withdrawal of consent to trial participation | |
| | | | 3.3.4.3 Discontinuation of the trial by the sponsor | |
| | | 3.3.5 | | |
| 4. | TRI | EATMI | ENTS | |
| •• | 4.1 | | STIGATIONAL TREATMENTS | |
| | 111 | 4.1.1 | Identity of the Investigational Medicinal Products | |
| | | 4.1.2 | Selection of doses in the trial | |
| | | 4.1.3 | Method of assigning subjects to treatment groups | |
| | | 4.1.4 | Drug assignment and administration of doses for each subject | |
| | | 4.1.5 | Blinding and procedures for unblinding | |
| | | 4.1.6 | Packaging, labelling, and re-supply | |
| | | 4.1.7 | Storage conditions | |
| | | 4.1.8 | Drug accountability | 30 |
| | 4.2 | OTHE | ER TREATMENTS, EMERGENCY PROCEDURES, | |
| | | REST | RICTIONS | 31 |
| | | 4.2.1 | Other treatments and emergency procedures | 31 |
| | | 4.2.2 | Restrictions | 31 |
| | | | 4.2.2.1 Restrictions regarding concomitant treatment | |
| | | | 4.2.2.2 Restrictions on diet and life style | |
| | 4.3 | TREA | TMENT COMPLIANCE | 32 |
| <b>5.</b> | ASS | SESSM | ENTS | 33 |
| | 5.1 | ASSES | SSMENT OF EFFICACY | 33 |
| | 5.2 | ASSES | SSMENT OF SAFETY | 33 |
| | | 5.2.1 | Physical examination | 33 |
| | | 5.2.2 | Vital signs | |
| | | 5.2.3 | Safety laboratory parameters | |
| | | 5.2.4 | Electrocardiogram | |
| | | 5.2.5 | Other safety parameters | 36 |
| | | 5.2.6 | Assessment of adverse events | 36 |
| | | | 5.2.6.1 Definitions of adverse events | 36 |

7.4

7.5

7.5.1

7.5.2

c32737758-02 Trial Protocol

**** 

| P | roprietary | confidential i | information © | 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies | 3 |
|---|---|---|---|---|---|
| | | | | 5.2.6.1.1 Adverse event | 36 |
| | | | | 5.2.6.1.2 Serious adverse event | |
| | | | | 5.2.6.1.3 AEs considered 'Always Serious' | 37 |
| | | | | 5.2.6.1.4 Adverse events of special interest | |
| | | | | 5.2.6.1.5 Intensity (severity) of AEs | |
| | | | | 5.2.6.1.6 Causal relationship of AEs | |
| | | | 5.2.6.2 | Adverse event collection and reporting | |
| | | | | 5.2.6.2.1 AE collection | |
| | | | | 5.2.6.2.2 AE reporting to the sponsor and timelines | |
| | | | | 5.2.6.2.3 Information required | 40 |
| | 5.3 | | | ENTRATION MEASUREMENTS AND | 40 |
| | | | | KINETICS | |
| | | 5.3.1 | | nent of pharmacokinetics | |
| | | 5.3.2 | | ls of sample collection | |
| | | | 5.3.2.1 | Blood sampling for pharmacokinetic analysis of BI 706321 | 40 |
| | 5.4 | RIOR | ANKINC | (<br> | 12 |
| | 5. <del>4</del> | | | SSMENTS | |
| | 5.6 | | | ENESS OF MEASUREMENTS | |
| | | | | NAL PLAN | |
| 6. | | | | | |
| | 6.1 | | | ULE | |
| | 6.2 | | | TRIAL PROCEDURES AT SELECTED VISITS | |
| | | 6.2.1 | | ng period | |
| | | 6.2.2 | | ent periods | |
| | | 6.2.3 | | up period and trial completion | |
| 7. | STA | TISTI | CAL M | ETHODS AND DETERMINATION OF | |
| | SAN | MPLE S | SIZE | | 45 |
| | 7.1 | STAT | ISTICAI | DESIGN – MODEL | 45 |
| | 7.2 | NULL | AND AI | LTERNATIVE HYPOTHESES | 45 |
| | 7.3 | | | ALYSES | |
| | | 7.3.1 | Primar | y endpoint analyses | 46 |
| | | 7.3.2 | | ary endpoint analyses | |

INTERIM ANALYSES ......48

HANDLING OF MISSING DATA ......48

Safety......48

c32737758-02 Trial Protocol 

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| | 7.6 | RANDOMISATION | 49 |
|---|---|---|---|
| | 7.7 | DETERMINATION OF SAMPLE SIZE | |
| 8. | INF | ORMED CONSENT, TRIAL RECORDS, DATA | |
| • | | OTECTION, PUBLICATION POLICY, AND | |
| | | MINISTRATIVE STRUCTURE | 51 |
| | 8.1 | TRIAL APPROVAL, SUBJECT INFORMATION, INFORMED | |
| | | CONSENT | 51 |
| | 8.2 | DATA QUALITY ASSURANCE | 52 |
| | 8.3 | RECORDS | 52 |
| | | 8.3.1 Source documents | 52 |
| | | 8.3.2 Direct access to source data and documents | 53 |
| | | 8.3.3 Storage period of records | 53 |
| | <b>8.4</b> | EXPEDITED REPORTING OF ADVERSE EVENTS | 53 |
| | 8.5 | STATEMENT OF CONFIDENTIALITY AND SUBJECT PRIVACY | 54 |
| | | 8.5.1 Collection, storage and future use of biological samples and corresponding data | 54 |
| | 8.6 | TRIAL MILESTONES | |
| | <b>8.7</b> | ADMINISTRATIVE STRUCTURE OF THE TRIAL | 55 |
| 9. | REI | FERENCES | 56 |
| | 9.1 | PUBLISHED REFERENCES | 56 |
| | 9.2 | UNPUBLISHED REFERENCES | |
| 10. | APF | PENDICES | 59 |
| 11. | DES | SCRIPTION OF GLOBAL AMENDMENT(S) | 60 |
| | | GLOBAL AMENDMENT 1 | |

Boehringer Ingelheim 01 Feb 2021

BI Trial No.: 1425-0010

c32737758-02 Trial Protocol 

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### **ABBREVIATIONS**

AE Adverse event

AESI Adverse events of special interest

ANOVA Analysis of variance

 $AUC_{0-\infty}$  Area under the concentration-time curve of the analyte in plasma over the

time interval from 0 extrapolated to infinity

 $AUC_{0-tz}$  Area under the concentration-time curve of the analyte in plasma over the

time interval from 0 to the last quantifiable data point

BA Bioavailability

BI Boehringer Ingelheim

BMI Body mass index (weight divided by height squared)

BP Blood pressure
bpm Beats per minute
CA Competent authority

CI Confidence interval

C<sub>max</sub> Maximum measured concentration of the analyte in plasma

CML Clinical Monitor Local

COVID-19 SARS-CoV-2 induced disease

CRF Case Report Form, paper or electronic (sometimes referred to as 'eCRF')

CTP Clinical trial protocol
CTR Clinical trial report

CV Arithmetic coefficient of variation

CYP Cytochrome P450
DDI Drug-drug interaction
DILI Drug induced liver injury

ECG Electrocardiogram

eCRF Electronic case report form eDC Electronic data capture

EDTA Ethylenediaminetetraacetic acid

EoTrial End of trial

EudraCT European Clinical Trials Database

01 Feb 2021

Boehringer Ingelheim BI Trial No.: 1425-0010

c32737758-02 Trial Protocol 

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

FIH First in Human FU Follow-up

GCP Good Clinical Practice

gCV Geometric coefficient of variation

IB Investigator's brochure ICF Informed Consent Form

IEC Independent Ethics CommitteeIPD Important protocol deviationIRB Institutional Review Board

ISF Investigator site file

LC-MS/MS Liquid chromatography with tandem mass spectrometry

LLOQ Lower Limit of Quantitation
MDA Methylenedioxyamphetamine
MDMA Methylenedioxymethamphetamine

MedDRA Medical Dictionary for Regulatory Activities

NOAEL No Observed Adverse Effect Level
NOD Nucleotide Oligomerization Domain

PCR Polymerase Chain Reaction

P-gp P-glycoprotein
PK Pharmacokinetic(s)
PKS Pharmacokinetic set

PMDA Pharmaceuticals and Medicinal Devices Agency

PR Pulse rate

q.d. Quaque die, once daily

QT Time between start of the Q-wave and the end of the T-wave in an

electrocardiogram

QT or or of the

or Bazett (QTcB)

R Reference treatment
REP Residual effect period

SAE Serious adverse event

SARS-CoV-2 Severe acute respiratory syndrome coronavirus 2

SCR Screening

SmPC Summary of Product Characteristics

SOP Standard operating procedure

**Boehringer Ingelheim** BI Trial No.: 1425-0010

c32737758-02

01 Feb 2021

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

**Trial Protocol** 

Single-rising dose SRD

Test product or treatment T

| | 1 |
|-------|----------------------------------------------------------------|
| TS | Treated set |
| $t_z$ | Time of last measurable concentration of the analyte in plasma |
| TSAP | Trial statistical analysis plan |
| ULN | Upper limit of normal |
| XTC | Ecstasy |


c32737758-02

Trial Protocol


Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 1. INTRODUCTION

#### 1.1 MEDICAL BACKGROUND



For more details on medical background refer to the Investigator's Brochure (IB) [c26475781].

#### 1.2 DRUG PROFILE

#### 1.2.1 BI 706321

For details on the nonclinical pharmacology, pharmacokinetics in animals and toxicology results refer to the IB [c26475781].

As of 28 May 2020, preliminary results are available from Part I of the <u>first-in-human Trial 1425-0001</u>. A total of 46 healthy male subjects received single oral ascending doses of BI 706321 and 15 subjects received placebo.

All tested doses of BI 706321 have been well tolerated. The observed AEs did not follow any specific pattern of distribution and no dose dependency was observed. Neither SAE nor severe AE were observed. The frequency of subjects with at least one treatment-emergent AE ranged from 0 to 60% on BI 706321 dose groups as compared to 40% on placebo. AEs reported in >1 subject on active treatment were coded as diarrhea (n=2, loose stool and watery stool and nasopharyngitis (n=2, loose stool dizziness). A total of 5 drug related AEs have been observed on active treatment: dry lips and loose stool dizziness




The "generalized sensation of cold" was accompanied by a slightly increased body temperature (37.4°C) and an increased CRP-value (35.4 mg/l). Beyond this no specific changes of laboratory parameters have been observed in the tested dose groups. Clinical monitoring did not show any relevant changes of ECG-parameters and vital signs [c26475781].



As of 21 September 2020, an additional 16 subjects were dosed with part of the blinded first and second dose cohorts of the multiple rising dose Trial 1425-0002. Both tested doses of BI 706321 were well-tolerated and neither SAE nor severe AE were observed.

#### 1.2.2 Itraconazole

Absorption of itraconazole solution is fast with maximum plasma concentration being reached within 2.5 h after oral administration in fasting condition. Bioavailability of itraconazole liquid increases by 30% when given under fasting condition compared to administration together with food [R20-2709]. Mean peak plasma concentrations were 547.7 ng/mL after a single dose of 200 mg itraconazole solution (fasting) and 1965 ng/mL after 15 days of daily treatment with 200 mg itraconazole solution (fasting). Pharmacokinetics of itraconazole is non-linear. The half-life of itraconazole after multiple doses of 200 mg once daily with solution formulation was about 40 h [R17-3742].

In the liver, itraconazole is metabolised extensively to more than 30 metabolites [R17-3743]. Its main metabolite, hydroxy-itraconazole, accounts for about twice the concentration of plasma itraconazole at trough. It has been shown *in vitro* that CYP3A4 is mainly responsible for the formation of this metabolite [R20-2709]. FDA classifies itraconazole as strong index inhibitor of CYP3A and as inhibitor of P-glycoprotein (P-gp) [R18-0241]. However, not only itraconazole contributes to the in vivo inhibition of CYP3A observed after itraconazole administration but also three of its metabolites (hydroxy-itraconazole, keto-itraconazole, and N desalkyl-itraconazole) [R10-1102].

For a more detailed description of itraconazole, please refer to the German Summary of Product Characteristics (SmPC) for Sempera<sup>®</sup> Liquid 10 mg/ml [R20-2709].

c32737758-02 Trial Protocol


Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 1.2.3 Residual Effect Period

The Residual Effect Period (REP, i.e., the period after the last dose with measurable drug levels and/or pharmacodynamic effects still likely to be present) of BI 706321 is assumed to be 8 days, i.e. based on  $\frac{1}{2}$  terminal  $t_{1/2}$  seen in the FIH trial 1425-0001.

When given together with itraconazole (Treatment T), it is expected that plasma exposure of BI 706321 could be increased (albeit within the exposures explored in the clinical trial 1425-0001), and the time of relevant plasma exposure could be prolonged. This might result in a prolonged period in which adverse effects could potentially occur.

For the use of itraconazole in Treatment T, the REP is defined as 8 days after last administration of itraconazole on Day 11 in Period 2.

#### 1.3 RATIONALE FOR PERFORMING THE TRIAL

Based on *in vitro* data, BI 706321 is mainly metabolized via CYP 3A4. Additionally, BI 706321 is an *in vitro* substrate of P-glycoprotein (P-gp).

Therefore, in this trial, the focus is on the drug-drug interaction (DDI) victim potential of BI 706321 with regard to CYP3A4 and P-gp as this may lead to clinically relevant increases in exposures with potential impact on patient safety.

Itraconazole is chosen for this trial as perpetrator drug, as this drug is recommended as strong inhibitor of CYP3A by EMA and PMDA [P15-06991, P15-06298], and as strong index inhibitor of CYP3A and P-gp by FDA [R18-0241].

Moreover, safety and tolerability of itraconazole were acceptable in previous DDI trials [c02336088, c03355329, c08928447].

#### 1.4 BENEFIT - RISK ASSESSMENT

Participation in this clinical trial is without any (therapeutic) benefit for healthy subjects. Their participation, however, is of major importance for the development of a drug which might improve the therapy of patients with Crohn's disease.

Subjects are exposed to risks of study procedures and risks related to the exposure to the trial medication.

#### 1.4.1 Procedure-related risks

The use of an indwelling venous catheter or venepuncture for e.g. blood sampling may result in mild bruising, and in rare cases, in transient inflammation of the wall of the vein, or nerve injury, potentially resulting in paraesthesia, reduced sensibility, and/or pain for an indefinite period, as well as in feeling of lightheadedness or in syncope.

The total volume of blood withdrawn per subject during the entire study will not exceed the volume of a normal blood donation (500 mL). No health-related risk to healthy subjects is expected from withdrawal of this volume of blood.

ECG electrodes may cause local and typically transient skin reactions.


Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 1.4.2 Drug-related risks and safety measures

#### 1.4.2.1 Drug induced liver injury

Although rare, a potential for drug-induced liver injury (DILI) is under constant surveillance by sponsors and regulators. Therefore, this trial requires timely detection, evaluation, and follow-up of laboratory alterations in selected liver laboratory parameters to ensure subjects' safety; see also Section 5.2.6.1.4, adverse events of special interest.

#### 1.4.2.2 BI 706321



### 1.4.2.2.1 Drug-related events observed in clinical trials with BI 706321

In Part I of the first-in-human trial 1425-0001, single ascending doses of BI 706321 have been well tolerated up to the maximum tested dose of [ref. Section 1.2.1].

Furthermore, multiple dose administration of q.d. over 14 days have been well tolerated in the first and second dose cohorts of the ongoing multiple rising dose trial 1425-0002.

As with all drugs, the potential for hypersensitivity and allergic reactions has to be taken into consideration when BI 706321 is administered.

#### 1.4.2.2.2 Risk assessment in the context of SARS-CoV-2 infection



Participation in this clinical trial will increase the risk of COVID-19 exposure due to traveling to the study site and completing the protocol-defined procedures at the study site. A risk management plan has been set up at the clinical site that detail specific precautionary measures, (e.g. hygiene rules, wearing of face masks, physical distancing), screening for SARS-CoV-2, and trial drug discontinuation in subjects with COVID-19 infection.


Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| 1.4.2.2.3 | Events predicted based on pharmacological properties / preclinical information |
|---|---|


Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies



#### 1.4.2.3 Itraconazole

In this trial, itraconazole will be used in a standard clinical dose of 200 mg once daily for 14 days. Multiple dosing of 200 mg itraconazole up to 15 days was of acceptable tolerability in healthy subjects [c02336088, c03355329, c08928447, R17-3742].

For a detailed description of the potential risks of itraconazole treatment in patients, please refer to the German Summary of Product Characteristics (SmPC) for Sempera<sup>®</sup> Liquid 10 mg/ml [R20-2709].

In order to address the risk of hepatotoxicity, only subjects with normal liver enzyme values will be included into the study. Safety laboratory parameters will be monitored closely. An individual subject will be removed from trial treatment if the subject shows an elevation of AST and/or ALT  $\geq$ 3-fold ULN combined with an elevation of total bilirubin  $\geq$ 2-fold ULN (measured in the same blood sample, see Section 3.3.4.1).

Further, most of the reported cases of serious hepatotoxicity during itraconazole treatment occurred in patients that suffered from concomitant liver diseases, had other significant diseases, or took concomitant hepatotoxic drugs. Subjects with liver diseases or a medical history of drug-induced liver failure are excluded from trial participation.

Itraconazole has shown a dose-related increase in maternal toxicity, embryotoxicity and teratogenicity in nonclinical studies at high doses, and therefore itraconazole must not be used during pregnancy. Woman of childbearing potential have to use a highly effective method of contraception until the menstrual period after the last itraconazole dose [R20-2709, R18-2643]. For risk mitigation, only male subjects will be included into this clinical trial.

Considering these safety measures and taking into account the reported acceptable tolerability of itraconazole, the planned administration of itraconazole does not represent an undue risk to healthy male volunteers.

#### 1.4.2.4 Potential drug-drug interaction between BI 706321 and itraconazole

It is likely that concomitant administration of BI 706321 with itraconazole leads to an increase of plasma concentrations and terminal half-live of BI 706321. The effect of itraconazole in increasing  $C_{max}$  and AUC of other drugs can be as high as 3.4-fold and 11-fold, respectively, as seen with oral midazolam, a sensitive CYP3A4 substrate, when coadministered with oral itraconazole 200 mg/d [R01-0516, R20-2709].

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Inhibition of P-gp may increase exposure of sensitive P-gp substrates like fexofenadine by factor 3-4 [R08-1652, P07-13746] and increase digoxin exposure by ~1.7-fold [R15-3252]. Therefore, a low dose of BI 706321 has been selected for this trial (see Section 4.1.2) to ensure that BI 706321 plasma concentrations, even in case of a substantial increase when given with itraconazole, are within the range of concentrations that were explored in the SRD part of trial 1425-0001 and that were associated with good safety and tolerability (ref. Section 1.2.1).

c32737758-02 Trial Protocol 

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## 2. TRIAL OBJECTIVES AND ENDPOINTS

#### 2.1 MAIN OBJECTIVES, PRIMARY AND SECONDARY ENDPOINTS

#### 2.1.1 Main objectives

The main objective of this trial is to investigate the effect on the exposure of BI 706321 in plasma when given as oral single dose together with multiple oral doses of itraconazole (Test, T) as compared to when given alone as oral single dose (Reference, R).

#### 2.1.2 Primary endpoints

The following pharmacokinetic parameters will be determined for BI 706321:

- AUC<sub>0- $\infty$ </sub> (area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity)
- C<sub>max</sub> (maximum measured concentration of the analyte in plasma)

#### 2.1.3 Secondary endpoint

The following pharmacokinetic parameter will be determined for BI 706321:

• AUC<sub>0-tz</sub> (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable data point)



Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies



## 2.2.2.2 Safety and tolerability

Safety and tolerability of the treatments will be assessed based on:

- Adverse events (including clinically relevant findings from the physical examination)
- Safety laboratory tests
- 12-lead ECG
- Vital signs (body temperature, blood pressure, pulse rate)

c32737758-02 Trial Protocol


Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 3. DESCRIPTION OF DESIGN AND TRIAL POPULATION

#### 3.1 OVERALL TRIAL DESIGN AND PLAN

The study will be performed as an open-label, two-treatment, two-period, fixed sequence design trial in healthy male subjects in order to compare the test treatment (T) to the reference treatment (R). The treatments will be one oral single dose of BI 706321 administered as tablet formulation together with multiple oral doses of 200 mg itraconazole as oral solution formulation (concentration: 10 mg/mL) (treatment T) and one single dose of BI 706321 as tablet given alone (R).

In both treatments, BI 706321 is administered to subjects in the fasting state. In the first treatment period (Period 1, Visit 2), all subjects are planned to undergo treatment R, and in the second treatment period (Period 2, Visit 3), all subjects are planned to undergo treatment T. For details, refer to Section 4.1.

There will be a washout period of at least 14 days between the administrations of BI 706321.



Figure 3.1: 1 Trial design

An overview of all relevant trial activities is provided in the <u>Flow Chart</u>. For visit schedule and details of trial procedures at selected visits, refer to Sections <u>6.1</u> and <u>6.2</u>, respectively.

## 3.2 DISCUSSION OF TRIAL DESIGN, INCLUDING THE CHOICE OF CONTROL GROUPS

For drug interaction trials, the crossover design is preferred because of its efficiency: since each subject serves as his/her own control, the comparison between treatments is based on an intra-subject comparison, thus removing inter-subject variability from the comparison between treatments [R94-1529].

Because of the long half-life (about 40 h) of itraconazole and its metabolites, a two-period fixed sequence design was selected, with administration of itraconazole in the second study period only. This design is not expected to lead to systematic errors in the estimation of the treatment effects since nonspecific time-effects are unlikely due to the short trial duration. For itraconazole studies, this design is recommended by the Innovation and Quality in


Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Pharmaceutical Development's 3744].

<u>[R17-</u>

For this PK drug-drug interaction trial, open-label treatment is acceptable, because the primary and secondary endpoints of this trial are PK endpoints derived from measurement of plasma concentrations of BI 706321. These endpoints are not expected to be affected by knowledge of treatment.

#### 3.3 SELECTION OF TRIAL POPULATION

It is planned that 14 healthy male subjects will enter the study. They will be recruited from the volunteers' pool of the trial site.

Due to the reproduction toxicity itraconazole has shown in nonclinical studies, only male subjects will be included in this trial.

A log of all subjects enrolled into the trial (i.e. who have signed informed consent) will be maintained in the ISF irrespective of whether they have been treated with investigational drug or not.

#### 3.3.1 Main diagnosis for trial entry

The study will be performed in healthy subjects.

#### 3.3.2 Inclusion criteria

Subjects will only be included in the trial if they meet the following criteria:

- 1. Healthy male subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (body temperature, BP, PR), 12-lead ECG, and clinical laboratory tests
- 2. Age of 18 to 50 years (inclusive)
- 3. BMI of 18.5 to 29.9 kg/m<sup>2</sup> (inclusive)
- 4. Signed and dated written informed consent prior to admission to the study, in accordance with GCP and local legislation

#### 3.3.3 Exclusion criteria

Subjects will not be allowed to participate, if any of the following general criteria apply:

- 1. Any finding in the medical examination (including BP, PR or ECG) deviating from normal and assessed as clinically relevant by the investigator
- 2. Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 45 to 90 bpm
- 3. Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
- 4. Any evidence of a concomitant disease assessed as clinically relevant by the investigator

c32737758-02


Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

- 5. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
- 6. Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair)
- 7. Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
- 8. History of relevant orthostatic hypotension, fainting spells, or blackouts
- 9. Relevant chronic or acute infections
- 10. History of relevant allergy or hypersensitivity (including allergy to the trial medication or its excipients)
- 11. Use of drugs within 30 days of planned administration of trial medication that might reasonably influence the results of the trial (including drugs that cause QT/QTc interval prolongation)
- 12. Intake of an investigational drug in another clinical trial within 60 days of planned administration of investigational drug in the current trial, or concurrent participation in another clinical trial in which investigational drug is administered
- 13. Smoker (more than 10 cigarettes or 3 cigars or 3 pipes per day)
- 14. Inability to refrain from smoking on specified trial days
- 15. Alcohol abuse (consumption of more than 24 g per day) and unwillingness/inability to refrain from intake of alcoholic beverages from 48 hours prior to first trial medication administration and until 7 days post last trial medication administration
- 16. Drug abuse or positive drug screening
- 17. Blood donation of more than 100 mL within 30 days of planned administration of trial medication or intended blood donation during the trial
- 18. Intention to perform excessive physical activities within one week prior to the administration of trial medication or during the trial
- 19. Inability to comply with the dietary regimen of the trial site
- 20. A marked prolongation of QT/QTc interval (such as QTc intervals that are repeatedly greater than 450 ms) or any other relevant ECG finding at screening
- 21. A history of additional risk factors for *Torsade de Pointes* (such as heart failure, hypokalaemia, or family history of Long QT Syndrome)
- 22. Subject is assessed as unsuitable for inclusion by the investigator, for instance, because the subject is not considered able to understand and comply with study requirements, or has a condition that would not allow safe participation in the study
- 23. Liver enzymes (ALT, AST, GGT) above upper limit of normal at the screening examination, confirmed by a repeat test
- 24. History of drug induced liver injury
- 25. History of heart failure, or any evidence of ventricular dysfunction
- 26. Known sorbitol/polyols intolerance
- 27. During COVID-19 pandemic: laboratory test indicative of an ongoing SARS-CoV-2 infection


Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

For study restrictions, refer to Section <u>4.2.2</u>.

### 3.3.4 Withdrawal of subjects from treatment or assessments

Subjects may discontinue trial treatment or withdraw consent to trial participation as a whole ('withdrawal of consent') with very different implications; please see sections <u>3.3.4.1</u> and <u>3.3.4.2</u> below.

If a subject is removed from or withdraws from the trial prior to the first administration of trial medication, the data of this subject will not be entered in the case report form (CRF) and will not be reported in the clinical trial report (CTR). If a subject is removed from or withdraws from the trial after the first administration of trial medication, this will be documented and the reason for discontinuation must be recorded in the CRF; in addition, the data will be included in the CRF and will be reported in the CTR. At the time of discontinuation, a complete end of trial examination will be performed, if possible, and the information will be recorded in the CRF. If the discontinuation occurs before the end of the REP (see Section 1.2.3), the discontinued subject should if possible be questioned for AEs and concomitant therapies at or after the end of the REP in order to ensure collection of AEs and concomitant therapies throughout the REP, if not contrary to any consent withdrawal of the subject.

#### 3.3.4.1 Discontinuation of trial treatment

An individual subject will discontinue trial treatment if:

- 1. The subject wants to discontinue trial treatment, without the need to justify the decision
- 2. The subject has repeatedly shown to be non-compliant with important trial procedures and, in the opinion of both, the investigator and sponsor representative, is not willing or able to adhere to the trial requirements in the future.
- 3. The subject needs to take concomitant medication that interferes with the investigational medicinal product or other trial treatment
- 4. The subject can no longer receive trial treatment for medical reasons (such as surgery, adverse events [AEs], or diseases)
- 5. An AE or clinically significant laboratory change or abnormality occurs that the investigator assesses as warranting discontinuation of treatment. This may include:
  - The subject has an elevation of AST and/or ALT ≥3-fold ULN
  - The subject has a serious adverse reaction or a severe non-serious adverse reaction
- 6. The subject has an elevation of AST and/or ALT ≥3-fold ULN <u>and</u> an elevation of total bilirubin ≥2-fold ULN (measured in the same blood sample) and/or needs to be followed up according to the DILI checklist provided in the ISF

In addition to these criteria, the investigator may discontinue subjects at any time based on his or her clinical judgment.

Even if the trial treatment is discontinued, the subject remains in the trial and, given his/her agreement, will undergo the procedures for early treatment discontinuation and follow up as outlined in the Flow Chart and section 6.2.3.

Trial Protocol 

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 3.3.4.2 Withdrawal of consent to trial participation

Subjects may withdraw their consent to trial participation at any time without the need to justify the decision. If a subject wants to withdraw consent, the investigator should be involved in the discussion with the subject and explain the difference between trial treatment discontinuation and withdrawal of consent to trial participation, as well as explain the options for continued follow up after trial treatment discontinuation, please see section 3.3.4.1 above

#### 3.3.4.3 Discontinuation of the trial by the sponsor

Boehringer Ingelheim reserves the right to discontinue the trial at any time for any of the following reasons:

- 1. Failure to meet expected enrolment goals overall or at a particular trial site
- 2. New toxicological findings, serious adverse events, or any safety information invalidating the earlier positive benefit-risk-assessment. More specifically, the trial will be terminated if more than 50% of the subjects have drug-related and clinically relevant adverse events of moderate or severe intensity, or if at least 1 drug-related serious adverse event is reported
- 3. Violation of GCP, or the CTP, or the contract with BI impairing the appropriate conduct of the trial
- 4. The sponsor decides to discontinue the further development of the investigational product

The investigator / trial site will be reimbursed for reasonable expenses incurred in case of trial termination (except if item 3 applies).

#### 3.3.5 Replacement of subjects

Subjects withdrawn due to drug related adverse events will not be replaced. In case more than 2 subjects do not complete the trial, the Clinical Trial Leader together with the Trial Pharmacokineticist and the Trial Statistician are to decide, if and how many subjects will be replaced. A replacement subject will be assigned a unique trial subject number.

c32737758-02 **Trial Protocol** 

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 4. **TREATMENTS**

#### 4.1 INVESTIGATIONAL TREATMENTS

The investigational product BI 706321 as tablet formulation will be supplied by BI Pharma GmbH & Co. KG.

Itraconazole oral solution will be obtained from a public pharmacy.

#### 4.1.1 **Identity of the Investigational Medicinal Products**

The characteristics of the trial products are given below:

Trial product 1

Substance: BI 706321

Pharmaceutical formulation: Tablet, film-coated

Source: BI Pharma GmbH & Co. KG, Germany

Unit strength:

1-0-0 Posology:

Route of administration: Oral

Duration of use: Single dose in treatments R and T

Trial product 2

Sempera® Liquid 10 mg/mL Name:

Itraconazole Substance:

Pharmaceutical formulation: Oral solution

Source: Public pharmacy

Holder of marketing

authorisation:

10 mg/mL

Unit strength: 20 mL-0-0 Posology:

Route of administration: Oral

Duration of use: 14 days in treatment T

#### 4.1.2 Selection of doses in the trial

#### Perpetrator (itraconazole)

The dose of itraconazole selected for this trial reflects standard clinical doses, is considered sufficient to yield significant CYP3A and P-gp inhibition and has been used successfully and safely in previous drug-drug-interaction trials (c02336088, c03355329, c08928447).

c32737758-02 Trial Protocol 

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### Victim (BI 706321)

Based on *in vitro* data, CYP3A is the major CYP isoform responsible for the metabolism of BI 706321. Additionally, BI 706321 is an *in vitro* substrate of P-gp. Thus, concomitant administration of BI 706321 with the strong CYP3A inhibitor itraconazole may result in substantial increases of BI 706321 plasma concentrations.

For the current trial, a dose of BI 706321 is selected, in order to ensure that BI 706321 plasma concentrations, even in case of a substantial increase when given with itraconazole, are within the range of concentrations that were explored in the SRD part of trial 1425-0001 and that were associated with good safety and tolerability (ref. Section 1.2.1).

#### 4.1.3 Method of assigning subjects to treatment groups

There is only one treatment sequence investigated in this trial, and each subject will be allocated to the same treatment sequence (R-T). The subjects will be allocated to a study subject number by the method "first come-first served" prior to first administration of trial medication in the morning of Day 1 of Visit 2. Once a subject number has been assigned, it cannot be reassigned to any other subject.

All subjects may be treated in one cohort, i.e. all subjects may receive treatment on the same calendar day. In case this is not feasible (e.g., due to logistical or recruitment reasons), the group may be split into several cohorts as required.

Treatment of all subjects on the same calendar day is acceptable (for safety margin to exposure reached in previous SRD trial 1425-0001 refer to Section 1.4.2.1.1; for discussion of study-associated risks and safety measures see Section 1.4).

#### 4.1.4 Drug assignment and administration of doses for each subject

The treatments to be evaluated are outlined in Table 4.1.4: 1 below. All subjects will receive the 2 treatments in a fixed order.

Table 4.1.4: 1 Dosage and treatment schedule

| Treatment period | Treatment | Substance | Formulation | Unit<br>strength | Dosage | Total<br>dose |
|---|---|---|---|---|---|---|
| 1 | R (Reference) | BI 706321 | Tablet, film-coated | | 1 tablet as single dose<br>(Day 1) | |
| 2 | T (Test) | BI 706321 | Tablet, film-coated | | 1 tablet as single dose<br>(Day 1) | |
| | | Itraconazole | Oral solution | 10 mg/mL | 20 mL (200 mg) qd for 14 days<br>(Days -3 to 11) | 2800 mg |

Administration of trial medication will be performed after subjects have fasted overnight; fasting is to start no later than 10 h before the scheduled dosing of BI 706321 or 9 hours before itraconazole administration. The investigator (or authorised designee) will administer the trial medication as an oral dose together with about 240 mL of water to subjects who are in a standing or sitting position. For drug administration, the so-called four-eye principle (two-person rule) should be applied. For this, one authorised employee of the trial site should

c32737758-02

**Trial Protocol** 


Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

witness the administration of trial medication, and – if applicable – its preparation (e.g. reconstitution), if correct dosage cannot be ensured otherwise.

Subjects will be kept under close medical surveillance until at least 24 hours and 46 hours after administration of BI 706321 in Visit 2 and Visit 3, respectively. During the first 4 h after administration of BI 706321, subjects are not allowed to lie down (i.e. no declination of the upper body of more than 45 degrees from upright posture).

The treatments with BI 706321 will be separated by a wash-out phase of at least 14 days.

## 4.1.5 Blinding and procedures for unblinding

This Phase I trial will be handled in an open fashion throughout (that is, during the conduct, including data cleaning and preparation of the analysis). This is considered acceptable because the potential for bias seems to be low and does not outweigh practical considerations.

Due to the open design of this trial, emergency envelopes will not be provided.

#### 4.1.6 Packaging, labelling, and re-supply

#### BI 706321

BI 706321 tablets will be provided by BI. They will be packaged and labelled in accordance with local law and the principles of Good Manufacturing Practice.

For details of packing and the description of the label, refer to the ISF.

The telephone number of the sponsor and the name, address and telephone number of the trial site are provided in the subject information form. The EudraCT number is indicated on the title page of this protocol as well as on the subject information and informed consent forms.

No re-supply is planned.

#### Itraconazole

Itraconazole oral solution will be obtained by the clinical trial site from a public pharmacy. The drug will be dispensed out of the original, unmodified packages.

#### 4.1.7 Storage conditions

Drug supplies will be kept in their original packaging and in a secure limited access storage area in accordance with the recommended (labelled) storage conditions. If necessary, a temperature log must be maintained to make certain that the drug supplies are stored at the correct temperature. If the storage conditions are found to be outside the specified range, the local clinical monitor (as provided in the list of contacts) is to be contacted immediately.

#### 4.1.8 Drug accountability

The investigator or designee will receive the investigational drugs delivered from the sponsor following requirements are fulfilled:

• Approval of the clinical trial protocol by the IRB / ethics committee

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

- Availability of a signed and dated clinical trial contract between the sponsor and the investigational site
- Approval/notification of the regulatory authority, e.g. competent authority
- Availability of the curriculum vitae of the Principal Investigator
- Availability of a signed and dated clinical trial protocol

Only authorised personnel documented in the form 'Trial Staff List' may dispense medication to trial subjects. The trial medication must be administered in the manner specified in the CTP.

The investigator or designee must maintain records of the product's delivery to the trial site, the inventory at the site, the use by each subject, and the disposal of unused products. These records will include dates, quantities, batch / serial numbers, expiry ('use-by') dates, and the unique code numbers assigned to the investigational medicinal product and trial subjects. The investigator or designee will maintain records that document adequately that the subjects were provided the doses specified by the CTP and reconcile all investigational medicinal products received from the sponsor. At the time of disposal of remaining trial medication, the investigator or designee must verify that no remaining supplies are in the investigator's possession.

All unused medication will be disposed of locally by the trial site upon written authorisation of the trial clinical monitor. Receipt, usage and disposal of trial medication must be documented on the appropriate forms. Account must be given for any discrepancies.

## 4.2 OTHER TREATMENTS, EMERGENCY PROCEDURES, RESTRICTIONS

#### 4.2.1 Other treatments and emergency procedures

There are no special emergency procedures to be followed. No additional treatment is planned. However, if adverse events require treatment, the investigator can authorise symptomatic therapy. In those cases, subjects will be treated as necessary and, if required, kept under supervision at the trial site or transferred to a hospital until all results of medical evaluations are acceptable.

#### 4.2.2 Restrictions

## 4.2.2.1 Restrictions regarding concomitant treatment

In principle, no concomitant therapy is allowed. All concomitant or rescue therapies will be recorded (including time of intake on study days) on the appropriate pages of the CRF.

Known inhibitors/inducers of CYP3A4 or P-gp activity, drugs with a known hepatotoxicity profile, drugs which are contraindicated to be co-administered with itraconazole [R20-2709] should be avoided during the entire study; if necessary, short term use of ibuprofen is acceptable.


Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 4.2.2.2 Restrictions on diet and life style

Poppy-seeds containing foods should not be consumed starting 3 days before the first drug administration in each treatment period, in order to avoid false-positive results in the drug-screen.

While admitted to the trial site, the subjects will be instructed not to consume any foods or drinks other than those provided by the staff. Standardised meals will be served at the times indicated in the <u>Flow Chart</u>. No food is allowed within 10 h before and for at least 4 h after intake of BI 706321. Subjects will be advised to not consume any food within 9 h before and 1 h after itraconazole administrations.

On Day 1, from 1 h before intake of BI 706321 (Period 1) or itraconazole (Period 2), respectively, fluid intake is restricted to the water administered with the drug, and an additional 240 mL of water at 2 h and 4 h post-dose (mandatory for all subjects). From lunch until 23 h post-dose BI 706321, total fluid intake is restricted to 3000 mL.

Grapefruits, Seville oranges (sour or bitter oranges) and their juices, and dietary supplements and products containing St. John's wort (*Hypericum perforatum*) are not permitted from 7 days before the first administration of trial medication in Period 1 until after the last PK sample of Period 2 is collected.

Alcoholic beverages are not permitted from 3 days before the first administration of trial medication in Period 1 until after the last PK sample in Period 2 is collected.

Methylxanthine-containing drinks or foods (such as coffee, tea, cola, energy drinks, or chocolate) are not allowed from 10 h before until 24 h after administration of BI 706321.

Smoking is not allowed during in-house confinement.

Excessive physical activity (such as competitive sport) should be avoided from 7 days before the first administration of trial medication until the end of trial examination.

Direct exposure to the sun or exposure to solarium radiation should be avoided during the entire study.

#### 4.3 TREATMENT COMPLIANCE

Compliance will be assured by administration of all trial medication in the study centre under supervision of the investigating physician or a designee. The measured plasma concentrations of trial medication will provide additional confirmation of compliance.

Subjects who are non-compliant (for instance, who do not appear for scheduled visits or violate trial restrictions) may be removed from the trial and the CRF will be completed accordingly (for further procedures, please see Section 3.3.4).

c32737758-02  Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### **5. ASSESSMENTS**

#### 5.1 ASSESSMENT OF EFFICACY

Not applicable.

#### 5.2 ASSESSMENT OF SAFETY

#### 5.2.1 Physical examination

At screening, the medical examination will include demographics, height and body weight, smoking and alcohol history (result not mandatory to be entered into CRF or to be reported), relevant medical history and concomitant therapy, review of inclusion and exclusion criteria, review of vital signs (body temperature, BP, PR), 12-lead ECG, laboratory tests, and a physical examination. At the end of trial examination, it will include review of vital signs, 12lead ECG, laboratory tests, and a physical examination.

#### 5.2.2 Vital signs

Systolic and diastolic blood pressures (BP) as well as pulse rate (PR) will be measured by a blood pressure monitor (Dinamap, indicated in the Flow Chart, after subjects have rested for at least 5 min in a supine position. All recordings should be made using the same type of blood pressure recording instrument on the same arm, if possible. Body temperature will be measured using ear thermometer.

#### 5.2.3 Safety laboratory parameters

For the assessment of laboratory parameters, blood and urine samples will be collected by the trial site at the times indicated in the Flow Chart after the subjects have fasted for at least 10 h. For retests, at the discretion of the investigator or designee, overnight fasting is not required.

The parameters that will be determined are listed in Tables 5.2.3: 1 and 5.2.3: 2. Reference ranges will be provided in the ISF.

Manual differential white blood cell count or urine sediment examinations will only be performed if there is an abnormality in the automatic blood cell count or in the urinalysis, respectively.

c32737758-02 Trial Protocol


Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## Table 5.2.3: 1 Routine laboratory tests

| Functional lab group | BI test name [comment/abbreviation] | A <sup>1</sup> | $\mathbf{B}^1$ | $\mathbf{C}^1$ | $\mathbf{D}^1$ |
|---|---|---|---|---|---|
| Haematology | Haematocrit | X | X | | X |
| | Haemoglobin | X | X | | X |
| | Red Blood Cell Count/Erythrocytes | X | X | | X |
| | Reticulocytes, absol. | X | X | | X |
| | Reticulocytes/Erythrocyte | X | X | | X |
| | White Blood Cells/Leukocytes | X | X | | X |
| | Platelet Count/Thrombocytes (quant) | X | X | | X |
| Automatic WBC | Neutrophils/Leukocytes; Eosinophils/Leukocytes; Basophils/ | | X | | X |
| differential, relative | Leukocytes; Monocytes/Leukocytes; Lymphocytes/Leukocytes | | | | |
| Automatic WBC | Neutrophil, absol.; Eosinophils, absol.; Basophils, absol.; | | X | | X |
| differential, absolute | Monocytes, absol.; Lymphocytes, absol. | | | | |
| Manual differential | Neut. Poly (segs)/Leukocytes; Neut. Poly (segs), absol.; Neutrophils | | | | |
| WBC (if automatic | Bands/Leukocytes; Neutrophils Bands, absol.; | | | | |
| differential WBC is | Eosinophils/Leukocytes; Eosinophils, absol.; Basophils/Leukocytes; | | | | |
| abnormal) | Basophils, absol.; Monocytes/Leukocytes; Monocytes, absol.; | | | | |
| | Lymphocytes/Leukocytes; Lymphocytes, absol. | | | | |
| Coagulation | Activated Partial Thromboplastin Time | X | | | X |
| | Prothrombin time | X | | | X |
| | INR (International Normalization Ratio) | X | | | X |
| | Fibrinogen | X | X | | X |
| Enzymes | AST [Aspartate transaminase] /GOT, SGOT | X | X | X | X |
| | ALT [Alanine transaminase] /GPT, SGPT | X | X | X | X |
| | Alkaline Phosphatase | X | X | X | X |
| | Gamma-Glutamyl Transferase) | X | X | X | X |
| | Creatine Kinase [CK] | X | X | | X |
| | Creatine Kinase Isoenzyme MB [only if CK is elevated] | X | X | | X |
| | Lactic Dehydrogenase | X | X | | X |
| Hormones | Thyroid Stimulating Hormone | X | | | |
| Substrates | Glucose (Plasma) | X | X | | X |
| | Creatinine | X | X | | X |
| | GFR/ CKD-EPI <sup>3</sup> | X | | | X |
| | Bilirubin, Total | X | X | X | X |
| | Bilirubin, Direct | X | X | X | X |
| | Protein, Total | X | X | | X |
| | C-Reactive Protein (Quant) | X | X | | X |
| | Haptoglobin | X | | | X |
| | Ferritin | X | | | X |
| | Cholesterol, total | X | | | X |
| Electrolytes | Sodium | X | X | | X |
| | Potassium | X | X | | X |
| Urinalysis <sup>2</sup> (Stix) | Urine Nitrite (qual) | X | | | X |
| | Urine Protein (qual) | X | | | X |
| | Urine Glucose (qual) | X | | | X |
| | Urine Ketone (qual) | X | | | X |
| | Urobilinogen (qual) | X | | | X |
| | Urine Bilirubin (qual) | X | | | X |
| | Urine RBC/Erythrocytes (qual) | X | | | X |
| | Urine WBC/Leucocytes (qual) | X | | | X |
| | Urine pH | X | | | X |
| Urine sediment <sup>2</sup> | Only positive findings will be reported (for instance, the presence of | | | | |
| Offile Sedifficial | | | | ı | 1 |
| Office sediment | sediment bacteria, casts in sediment, squamous epithelial cells, | | | | |


Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

- A: parameters to be determined at Visit 1 (screening examination)
  - B: parameters to be determined at Visit 2 and 3 (for study days and time points refer to Flow Chart)
  - C: parameters to be determined at Visit 3 (for study days and time points refer to Flow Chart)
  - D: parameters to be determined at Visit 4 (end of trial examination)
- <sup>2</sup> Microscopic examination if erythrocytes, leukocytes, nitrite or protein in urinalysis are abnormal in urine
- <sup>3</sup> Estimated glomerular filtration rate according to CKD-EPI formula (R12-1392)

The tests listed in Table <u>5.2.3: 2</u> are exclusionary laboratory tests that may be repeated as required. The results will not be entered in the CRF/database and will not be reported in the CTR. Except for drug screening, it is planned to perform these tests during screening only. Drug screening will be performed at screening and prior to first dose in each treatment period.

Depending on development of COVID-19 pandemic, testing for SARC-CoV-2 infection will be done (e.g. PCR) prior to inclusion into the study and may be repeated as deemed appropriate.

Table 5.2.3: 2 Exclusionary laboratory tests

| Functional lab group | Test name |
|---|---|
| Drug screening (urine) | Amphetamine/MDA Barbiturates Benzodiazepine Cannabis Cocaine Methadone Methamphetamines/MDMA/XTC Opiates |
| | Phencyclidine Tricyclic antidepressants |
| Infectious serology (blood) | Hepatitis B surface antigen (qualitative) Hepatitis B core antibody (qualitative) Hepatitis C antibodies (qualitative) HIV-1 and HIV-2 antibody (qualitative) |

To encourage compliance with alcoholic restrictions, a breath alcohol test (e.g. Alcotest® will be performed prior to each treatment period, and may be repeated at any time during the study at the discretion of an investigator or designee. The results will not be included in the CTR.

The laboratory tests listed in Tables <u>5.2.3: 1</u> and <u>5.2.3: 2</u> will be performed at

with the

exception of drug screening tests. These tests will be performed at the trial site using SureStep<sup>TM</sup> Multi-Drug Test (

Laboratory data will be transmitted electronically from the laboratory to the trial site.

c32737758-02 Trial Protocol


Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 5.2.4 Electrocardiogram

Twelve-lead ECGs (I, II, III, aVR, aVL, aVF, V1 - V6) will be recorded using a computerised electrocardiograph (CardioSoft EKG System, at the times provided in the Flow Chart.

To achieve a stable heart rate at rest and to assure high quality recordings, the site personnel will be instructed to assure a relaxed and quiet environment, so that all subjects are at complete rest.

All ECGs will be recorded for a 10 sec duration after subjects have rested for at least 5 min in a supine position. ECG assessment will always precede all other study procedures scheduled for the same time to avoid compromising ECG quality.

All ECGs will be stored electronically on the Muse CV Cardiology System (
Electrode placement will be performed according to the method of Wilson, Goldberger and Einthoven modified by Mason and Likar (hips and shoulders instead of ankles and wrists).

All locally printed ECGs will be evaluated by the investigator or a designee. Abnormal findings will be reported as AEs (during the trial) or baseline conditions (at screening) if assessed to be clinically relevant by the investigator. Any ECG abnormalities will be carefully monitored and, if necessary, the subject will be removed from the trial and will receive the appropriate medical treatment.

ECGs may be repeated for quality reasons (for instance, due to alternating current artefacts, muscle movements, or electrode dislocation) and the repeated ECG will be used for analysis. Additional (unscheduled) ECGs may be collected by the investigator for safety reasons.

#### 5.2.5 Other safety parameters

Not applicable.

#### 5.2.6 Assessment of adverse events

5.2.6.1 Definitions of adverse events

#### 5.2.6.1.1 Adverse event

An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation subject administered a medicinal product and which does not necessarily have to have a causal relationship with this treatment.

An AE can therefore be any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.

The following should also be recorded as an AE in the CRF and BI SAE form (if applicable):

• Worsening of the underlying disease or of other pre-existing conditions
Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

• Changes in vital signs, ECG, physical examination, and laboratory test results, if they are judged clinically relevant by the investigator

If such abnormalities already pre-exist prior to trial inclusion, they will be considered as baseline conditions and should be collected in the eCRF only.

#### 5.2.6.1.2 Serious adverse event

A serious adverse event (SAE) is defined as any AE which fulfils at least one of the following criteria:

- Results in death
- Is life-threatening, which refers to an event in which the patient was at risk of death at the time of the event; it does not refer to an event that hypothetically might have caused death if more severe
- Requires inpatient hospitalisation
- Requires prolongation of existing hospitalisation
- Results in persistent or significant disability or incapacity
- Is a congenital anomaly/birth defect
- Is deemed serious for any other reason if it is an important medical event when based upon appropriate medical judgment which may jeopardise the patient and may require medical or surgical intervention to prevent one of the other outcomes listed in the above definitions. Examples of such events are intensive treatment in an emergency room or at home for allergic bronchospasm, blood dyscrasias or convulsions that do not result in hospitalisation or development of dependency or abuse

#### 5.2.6.1.3 AEs considered 'Always Serious'

Cancers of new histology and exacerbations of existing cancer must be classified as a serious event regardless of the time since discontinuation of the trial medication and must be reported as described in <u>5.2.6.2</u>, subsections 'AE Collection' and 'AE reporting to sponsor and timelines'.

In accordance with the European Medicines Agency initiative on Important Medical Events, Boehringer Ingelheim has set up a list of further AEs, which, by their nature, can always be considered to be 'serious' even though they may not have met the criteria of an SAE as defined above.

The latest list of 'Always Serious AEs' can be found in the eDC system, an electronic data capture system which allows the entry of trial data at the trial site. These events should always be reported as SAEs as described above.

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 5.2.6.1.4 Adverse events of special interest

The term adverse events of special interest (AESI) relates to any specific AE that has been identified at the project level as being of particular concern for prospective safety monitoring and safety assessment within this trial, e.g. the potential for AEs based on knowledge from other compounds in the same class. AESIs need to be reported to the sponsor's Pharmacovigilance Department within the same timeframe that applies to SAEs, please see Section 5.2.6.2.2.

The following are considered as AESIs:

# Hepatic injury

A hepatic injury is defined by the following alterations of hepatic laboratory parameters:

- o An elevation of AST (aspartate transaminase) and/or ALT (alanine transaminase) ≥3-fold ULN combined with an elevation of total bilirubin ≥2-fold ULN measured in the same blood sample, or
- o Aminotransferase (ALT, and/or AST) elevations ≥10 fold ULN

These lab findings constitute a hepatic injury alert and the subjects showing these lab abnormalities need to be followed up according to the 'DILI checklist' provided in the ISF. In case of clinical symptoms of hepatic injury (icterus, unexplained encephalopathy, unexplained coagulopathy, right upper quadrant abdominal pain, etc.) without lab results (ALT, AST, total bilirubin) available, the Investigator should make sure that these parameters are analysed, if necessary in an unscheduled blood test. Should the results meet the criteria of hepatic injury alert, the procedures described in the DILI checklist should be followed.

#### 5.2.6.1.5 Intensity (severity) of AEs

The intensity (severity) of the AE should be judged based on the following:

Mild: Awareness of sign(s) or symptom(s) that is/are easily tolerated Moderate: Sufficient discomfort to cause interference with usual activity

Severe: Incapacitating or causing inability to work or to perform usual activities

### 5.2.6.1.6 Causal relationship of AEs

Medical judgment should be used to determine the relationship, considering all relevant factors, including pattern of reaction, temporal relationship, de-challenge or re-challenge, confounding factors such as concomitant medication, concomitant diseases and relevant history.

Arguments that may suggest that there is a reasonable possibility of a causal relationship could be:

- The event is consistent with the known pharmacology of the drug
- The event is known to be caused by or attributed to the drug class
- A plausible time to onset of the event relative to the time of drug exposure

c32737758-02


Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

- Evidence that the event is reproducible when the drug is re-introduced
- No medically sound alternative aetiologies that could explain the event (e.g. preexisting or concomitant diseases, or co-medications)
- The event is typically drug-related and infrequent in the general population not exposed to drugs (e.g. Stevens-Johnson syndrome)
- An indication of dose-response (i.e. greater effect size if the dose is increased, smaller effect size if dose is reduced)

Arguments that may suggest that there is no reasonable possibility of a causal relationship could be:

- No plausible time to onset of the event relative to the time of drug exposure is evident (e.g. pre-treatment cases, diagnosis of cancer or chronic disease within days / weeks of drug administration; an allergic reaction weeks after discontinuation of the drug concerned)
- Continuation of the event despite the withdrawal of the medication, taking into account the pharmacological properties of the compound (e.g. after 5 half-lives). Of note, this criterion may not be applicable to events whose time course is prolonged despite removing the original trigger
- Additional arguments amongst those stated before, like alternative explanation (e.g. situations where other drugs or underlying diseases appear to provide a more likely explanation for the observed event than the drug concerned)
- Disappearance of the event even though the trial drug treatment continues or remains unchanged

#### 5.2.6.2 Adverse event collection and reporting

#### 5.2.6.2.1 AE collection

Upon enrolment into a trial, the subject's baseline condition is assessed (for instance, by documentation of medical history/concomitant diagnoses), and relevant changes from baseline are noted subsequently.

Subjects will be required to report spontaneously any AEs as well as the time of onset, end time, and intensity of these events. In addition, each subject will be regularly assessed by the medical staff throughout the clinical trial and whenever the investigator deems necessary. As a minimum, subjects will be questioned for AEs (and concomitant therapies) at the time points indicated in the <u>Flow Chart</u>. Assessment will be made using non-specific questions such as 'How do you feel?'. Specific questions will be asked wherever necessary in order to more precisely describe an AE.

A carefully written record of all AEs shall be kept by the investigator in charge of the trial. Records of AEs shall include data on the time of onset, end time, intensity of the event, and any treatment or action required for the event and its outcome.

The following must be collected and documented on the appropriate CRF(s) by the investigator:

• From signing the informed consent onwards until an individual subject's end of trial:

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

All AEs (serious and non-serious) and all AESIs

Trial Protocol

The only exception to this rule are AEs (serious and non-serious) and AESIs in Phase I trials in healthy volunteers, when subjects discontinue from the trial due to screening failures prior to administration of any trial medication. In these cases, the subjects' data must be collected at trial site but will not be entered in the CRF or trial database and will not be reported in the CTR.


After the individual subject's end of trial:

c32737758-02

The investigator does not need to actively monitor the subject for AEs but should only report any occurrence of cancer and related SAEs and related AESIs of which the investigator may become aware of by any means of communication, e.g. phone call. Those AEs should, however, not be reported in the CRF.

#### AE reporting to the sponsor and timelines 5.2.6.2.2

The Investigator must report SAEs, AESIs, and non-serious AEs which are relevant for the reported SAE or AESI, on the BI SAE form immediately (within 24 hours) to the sponsor's unique entry point (country specific contact details will be provided in the ISF). The same timeline applies if follow-up information becomes available. In specific occasions the Investigator could inform the sponsor upfront via telephone. This does not replace the requirement to complete and send the BI SAE form.

With receipt of any further information to these events, a follow-up SAE form has to be provided. For follow-up information, the same rules and timeline apply as for initial information.

#### 5.2.6.2.3 Information required

All (S)AEs, including those persisting after the individual subject's end of trial, must be followed up until they have resolved, have been sufficiently assessed as 'chronic' or 'stable', or no further information can be obtained.

#### DRUG CONCENTRATION MEASUREMENTS AND 5.3 **PHARMACOKINETICS**

#### 5.3.1 **Assessment of pharmacokinetics**

For the assessment of pharmacokinetics, blood samples will be collected at the time points indicated in the Flow Chart. The actual sampling times will be recorded and used for determination of pharmacokinetic parameters.

#### 5.3.2 Methods of sample collection

#### 5.3.2.1 Blood sampling for pharmacokinetic analysis of BI 706321

For quantification of BI 706321 concentrations in plasma, 2.7 mL of blood will be drawn from an antecubital or forearm vein into an K2-EDTA (dipotassium


Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

ethylenediaminetetraacetic acid)-anticoagulant blood drawing tube at the times indicated in the <u>Flow Chart</u>. Blood will be withdrawn by means of either an indwelling venous catheter or by venepuncture with a metal needle.

The EDTA-anticoagulated blood samples will be centrifuged for approximately 10 min at approximately 2000 g to 4000 g and at 4 to 8 °C. Two plasma aliquots will be obtained and stored in polypropylene tubes. The first aliquot should contain at least 0.5 mL of plasma. The second aliquot should contain the remaining plasma.

The process from blood collection until transfer of plasma aliquots into the freezer should be completed within 60 min, with interim storage of blood samples in ice water or on ice. The time each aliquot was placed in the freezer will be documented. Until transfer on dry ice to the analytical laboratory, the aliquots will be stored upright at approximately -20°C or below at the trial site. The second aliquot will be transferred to the analytical laboratory after the bioanalyst has acknowledged safe arrival of the first aliquot. At the analytical laboratory, the plasma samples will be stored at approximately -20°C or below until analysis.

At a minimum, the sample tube labels should list BI trial number, subject number, visit, planned sampling time, and the analyte 'BI 706321'.



c32737758-02

Trial Protocol


Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies



#### 5.4 BIOBANKING

Not applicable.

#### 5.5 OTHER ASSESSMENTS

Not applicable.

#### 5.6 APPROPRIATENESS OF MEASUREMENTS

All measurements performed during this trial are standard measurements and will be performed in order to monitor subjects' safety and to determine pharmacokinetic parameters in an appropriate way. The scheduled measurements will allow monitoring of changes in vital signs, standard laboratory values, and ECG parameters that might occur as a result of administration of trial medication. The safety assessments are standard, are accepted for evaluation of safety and tolerability of an orally administered drug, and are widely used in clinical trials. The pharmacokinetic parameters and measurements outlined in Section <u>5.3</u> are generally used assessments of drug exposure.

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 6. INVESTIGATIONAL PLAN

#### 6.1 VISIT SCHEDULE

Exact times of measurements outside the permitted time windows will be documented. The acceptable time windows for screening, the end of trial examination, and measurements and assessments scheduled to occur 'before' trial medication administrations are provided in the Flow Chart.

If not stated otherwise in the Flow Chart, the acceptable deviation from the scheduled time for the assessment of safety (e.g. vital signs, ECG, laboratory tests) will be  $\pm$  30 min.

If scheduled in the Flow Chart at the same time as a meal, blood sampling, vital signs, and 12-lead ECG recordings have to be done first. Furthermore, if several measurements including venepuncture are scheduled for the same time, venepuncture should be the last of the measurements due to its inconvenience to the subject and possible influence on physiological parameters.

For planned blood sampling times, refer to the Flow Chart. While these nominal times should be adhered to as closely as possible, the actual sampling times will be recorded and used for the determination of pharmacokinetic parameters.

If a subject misses an appointment, it will be rescheduled if possible. The relevance of measurements outside the permitted time windows will be assessed no later than at the Report Planning Meeting.

#### 6.2 DETAILS OF TRIAL PROCEDURES AT SELECTED VISITS

#### 6.2.1 Screening period

After having been informed about the trial, all subjects will provide written informed consent in accordance with GCP and local legislation prior to enrolment in the study.

For information regarding laboratory tests (including drug and virus screening), ECG, vital signs, and physical examination, refer to Sections <u>5.2.1</u> to <u>5.2.4</u>.

## **6.2.2** Treatment periods

Each subject is expected to participate in 2 treatment periods (Day -3 to 9 in period 1 and Day -3 to 24 in period 2). At least 14 days will separate drug administration of BI 706321 in the first and second treatment period.

On Day 1 of each treatment period, study participants will be admitted to the trial site and kept under close medical surveillance for at least 24 h following drug administration in period 1 and for at least 46 hours following administration of BI 706321 in period 2. The subjects will then be allowed to leave the trial site after formal assessment and confirmation of their fitness. On all other study days, subjects will be treated in an ambulatory fashion.

For details on time points and procedures for collection of plasma samples for PK analysis, refer to Flow Chart and Section <u>5.3.2</u>.

Trial Protocol 

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

The safety measurements performed during the treatment period are specified in Section <u>5.2</u> of this protocol and in the <u>Flow Chart</u>. For details on times of all other trial procedures, refer to the Flow Chart. AEs and concomitant therapy will be assessed continuously from screening until the end of trial examination.

#### 6.2.3 Follow-up period and trial completion

For AE assessment, laboratory tests, recording of ECG and vital signs, and physical examination during the follow-up period, see Sections <u>5.2.1</u> to <u>5.2.6</u>. Subjects who discontinue treatment before the end of the planned treatment period should undergo the EoTrial Visit.

All abnormal values (including laboratory parameters) that are assessed as clinically relevant by the investigator will be monitored using the appropriate tests until a return to a medically acceptable level is achieved. (S)AEs persisting after a subject's EoTrial Visit must be followed until they have resolved, have been sufficiently characterised, or no further information can be obtained.

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 7. STATISTICAL METHODS AND DETERMINATION OF SAMPLE SIZE

#### 7.1 STATISTICAL DESIGN – MODEL

The main objective of this trial is to investigate the pharmacokinetics of BI 706321 in plasma when given as oral single dose together with multiple doses of itraconazole (Test, T) as compared to when given alone as oral single dose (Reference, R) on the basis of the primary and secondary pharmacokinetic endpoints, as listed in Sections 2.1.2 and 2.1.3. The trial is designed to allow intra-subject comparisons and will be evaluated statistically by use of a linear model for logarithmically transformed PK endpoints.

The assessment of safety is a further objective of this trial, and will be evaluated by descriptive statistics for the parameters specified in Section 2.2.2.2.

#### 7.2 NULL AND ALTERNATIVE HYPOTHESES

The relative bioavailability of BI 706321 given in combination with itraconazole (T) compared with BI 706321 given alone (R) will be estimated by the ratios of the geometric means (T/R), and their corresponding 2-sided 90% confidence intervals (CIs) will be provided. This method corresponds to the two one-sided t-test procedure, each at the 5% significance level. Since the main focus is on estimation and not testing, a formal hypothesis test and associated acceptance range is not specified.

#### 7.3 PLANNED ANALYSES

#### Analysis sets

Statistical analyses will be based on the following analysis sets:

- Treated set (TS): The treated set includes all subjects who were treated with at least one dose of study drug. The treated set will be used for safety analyses.
- Pharmacokinetic parameter analysis set (PKS): This set includes all subjects in the treated set (TS) who provide at least one PK endpoint that was defined as primary or secondary and was not excluded due to a protocol deviation relevant to the evaluation of PK or due to PK non-evaluability (as specified in the following subsection 'Pharmacokinetics'). Thus, a subject will be included in the PKS, even if he/she contributes only one PK parameter value for one period to the statistical assessment. Descriptive and model based analyses of PK parameters will be based on the PKS.

Adherence to the protocol will be assessed by the trial team. Important protocol deviation (IPD) categories will be suggested in the IPD specification file prior to trial initiation, IPDs will be identified no later than in the Report Planning Meeting, and the IPD categories will be updated as needed.


Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### Pharmacokinetics

The pharmacokinetic parameters listed in Section 2.1 for BI 706321 will be calculated according to the sponsor's SOP 'Standards and processes for analyses performed within Clinical Pharmacokinetics/ Pharmacodynamics' (001-MCS-36-472).

Plasma concentration data and parameters of a subject will be included in the statistical pharmacokinetic (PK) analyses if they are not flagged for exclusion due to a protocol deviation relevant to the evaluation of PK (to be decided no later than in the Report Planning Meeting) or due to PK non-evaluability (as revealed during data analysis, based on the criteria specified below). Exclusion of a subject's data will be documented in the CTR.

Relevant protocol deviations may be

- Incorrect trial medication taken, i.e. the subject received at least one dose of trial medication the subject was not assigned to
- Incorrect dose of trial medication taken
- Use of restricted medications

Plasma concentrations and/or parameters of a subject will be considered as non-evaluable, if for example

- The subject experienced emesis that occurred at or before two times median t<sub>max</sub> of the respective treatment (median t<sub>max</sub> is to be determined excluding the subjects experiencing emesis)
- A predose concentration of BI 706321 is >5% C<sub>max</sub> value of that subject in the respective treatment period
- Missing samples/concentration data at important phases of PK disposition curve

Plasma concentration data and parameters of a subject which is flagged for exclusion will be reported with its individual values but will not be included in the statistical analyses. Descriptive and inferential statistics of PK parameters will be based on the PKS.

Only concentration values within the validated concentration range and actual sampling times will be used for the calculation of pharmacokinetic parameters. Concentrations used in the pharmacokinetic calculations will be in the same format provided in the bioanalytical report, (that is, to the same number of decimal places provided in the bioanalytical report).

#### 7.3.1 Primary endpoint analyses

#### Primary analyses

The statistical model used for the analysis of the primary endpoints will be an analysis of variance (ANOVA) model on the logarithmic scale. That is, the PK endpoints will be log-transformed (natural logarithm) prior to fitting the ANOVA model. This model will include effects accounting for the following sources of variation: subjects and treatment. The effect 'subjects' will be considered as random, whereas 'treatment' will be considered as fixed. The model is described by the following equation:

$$y_{km} = \mu + s_m + \tau_k + e_{km}$$
, where

c32737758-02


Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

 $y_{km}$  = logarithm of response measured on subject m receiving treatment k,

 $\mu$  = the overall mean,

 $s_m$  = the effect associated with the m<sup>th</sup> subject, m = 1, 2, ..., n

 $\tau_k$  = the  $k^{th}$  treatment effect, k = 1, 2

 $e_{km} = \text{the random error associated with the } m^{th} \text{ subject who received treatment } k$  where  $s_m \sim N(0, \sigma_B^2) \text{ i.i.d.}, e_{km} \sim N(0, \sigma_W^2) \text{ i.i.d.}$  and  $s_m$ ,  $e_{km}$  are independent random variables.

Point estimates for the ratios of the geometric means (test/reference) for the primary endpoints (see Section 2.1) and their two-sided 90% confidence intervals (CIs) will be provided.

For each endpoint, the difference between the expected means for log(T)-log(R) will be estimated by the difference in the corresponding adjusted means (Least Squares Means). Additionally their two-sided 90% confidence intervals will be calculated based on the residual error from the ANOVA and quantiles from the t-distribution. These quantities will then be back-transformed to the original scale to provide the point estimate and 90% CIs for each endpoint.

#### Further exploratory analyses

The same statistical model as stated above will be repeated for the primary endpoints but with 'subjects' considered as fixed effects.

In addition to the model based approach all parameters will be calculated and analysed descriptively.

#### 7.3.2 Secondary endpoint analyses

The secondary endpoints (refer to Section 2.1.3) will be calculated according to the BI SOP 001-MCS-36-472 and will be assessed statistically using the same methods as described for the primary endpoints.



## 7.3.4 Safety analyses

Safety will be analysed based on the assessments described in Section <u>2.2.2.2</u>. All treated subjects (TS, refer to Section <u>7.2</u>) will be included in the safety analysis. Safety analyses will be descriptive in nature and based on BI standards. No hypothesis testing is planned.


Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

For all analyses, the treatment actually administered (= treatment at onset) to the subject will be used (any deviations from treatment will be discussed in the minutes of the Report Planning Meeting).

Treatments will be compared in a descriptive way. Tabulations of frequencies/proportions will be used to evaluate categorical (qualitative) data, and tabulations of descriptive statistics will be used to analyse continuous (quantitative) data.

Measurements (such as ECG, vital signs, or laboratory parameters) or AEs will be assigned to treatments (see Section 4.1) based on the actual treatment at the planned time of the measurement or on the recorded time of AE onset (concept of treatment emergent AEs). Therefore, measurements planned or AEs recorded prior to first intake of trial medication will be assigned to the screening period, those between first trial medication intake and end of REP (see Section 1.2.3) will be assigned to the treatment period. Events occurring after the REP but prior to next intake or end of trial termination date will be assigned to 'follow-up'. In case of two or more treatments, the follow-up will be summarized according to the previous treatment. These assignments including the corresponding time intervals will be defined in detail in the TSAP. Note that AEs occurring after the last per protocol contact but entered before final database lock will be reported to Pharmacovigilance only and will not be captured in the trial database.

Additionally, further treatment intervals (analysing treatments) may be defined in the TSAP in order to provide summary statistics for time intervals, such as combined treatments, ontreatment totals, or periods without treatment effects (such as screening and follow-up intervals).

Adverse events will be coded using the Medical Dictionary for Regulatory Activities (MedDRA). Frequency, severity, and causal relationship of AEs will be tabulated by treatment, system organ class, and preferred term. SAEs, AESIs (see Section <u>5.2.6.1</u>), and other significant AEs (according to ICH E3) will be listed separately.

Previous and concomitant therapies will be presented per treatment group without consideration of time intervals and treatment periods.

Laboratory data will be compared to their reference ranges. Values outside the reference range as well as values defined as possibly clinically significant will be highlighted in the listings. Additionally, differences from baseline will be evaluated.

Vital signs or other safety-relevant data will be assessed with regard to possible on-treatment changes from baseline.

#### 7.4 INTERIM ANALYSES

No interim analysis is planned.

#### 7.5 HANDLING OF MISSING DATA

#### **7.5.1** Safety

It is not planned to impute missing values for safety parameters.


Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 7.5.2 Pharmacokinetics

Handling of missing PK data will be performed according to the relevant Corporate Procedure (001-MCS-36-472).

PK parameters that cannot be reasonably calculated based on the available drug concentration-time data will not be imputed.

#### 7.6 RANDOMISATION

In this trial subjects receive all treatments in the same order, thus no randomisation for the treatment assignment is performed (see also Section 4.1.3).

#### 7.7 DETERMINATION OF SAMPLE SIZE

It is planned to enter a total of 14 subjects in the trial (accounting for up to 2 dropouts or non PK evaluable subjects), because this sample size is considered sufficient to achieve the aims of this exploratory trial. With this sample size, the following precision in estimating the ratio of geometric means (test/reference) can be expected with 95% probability. Precision is defined as the ratio of upper confidence interval (CI) limit to the estimate of ratio of geometric means. Note that the precision is independent of the actual ratio of geometric means.




Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Table 7.7: 1 Precision that can be expected with 95% probability and illustrative two-sided 90% confidence intervals around the ratios of geometric means (T/R) for different gCVs in a two-period fixed sequence trial (N=12)

| | Precision upper<br>CI limit / relative<br>BA estimate | Ratio [%]* | Lower CI limit<br>[%] | Upper CI limit<br>[%] |
|---|---|---|---|---|
| 20.0 | 1.21 | 100 | 82.35 | 121.43 |
| 20.0 | 1.21 | 150 | 123.53 | 182.15 |
| 20.0 | 1.21 | 200 | 164.70 | 242.86 |
| 25.0 | 1.27 | 100 | 78.55 | 127.31 |
| 25.0 | 1.27 | 150 | 117.83 | 190.96 |
| 25.0 | 1.27 | 200 | 157.10 | 254.61 |
| 30.0 | 1.33 | 100 | 74.99 | 133.36 |
| 30.0 | 1.33 | 150 | 112.48 | 200.03 |
| 30.0 | 1.33 | 200 | 149.98 | 266.71 |

<sup>\*</sup>Ratio of geometric means (test/reference) for a PK endpoint is defined by  $\exp(\mu_T)/\exp(\mu_R)$ .

The expected 90% confidence interval limits in the table were derived by

CI limit<sub>upper,lower</sub> = 
$$exp(ln(\theta) \pm \omega)$$
,

with  $\theta$  being the ratio (T/R) on original scale and  $\omega$  the distance from the estimate  $\theta$  to either confidence interval limit on the log-scale, which was obtained from the achievable precision on the original scale.

The calculation was performed as described by Julious [R11-5230] using R Version 3.6.1.

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 8. INFORMED CONSENT, TRIAL RECORDS, DATA PROTECTION, PUBLICATION POLICY, AND ADMINISTRATIVE STRUCTURE

Trial Protocol

c32737758-02

The trial will be carried out in compliance with the protocol, the ethical principles laid down in the Declaration of Helsinki, in accordance with the ICH Harmonized Guideline for Good Clinical Practice (GCP), relevant BI Standard Operating Procedures (SOPs), the EU regulation 536/2014, and other relevant regulations. Investigators and site staff must adhere to these principles.

Standard medical care (prophylactic, diagnostic, and therapeutic procedures) remains the responsibility of the subject's treating physician.

The investigator will inform the sponsor immediately of any urgent safety measures taken to protect the trial subjects against any immediate hazard, as well as of any serious breaches of the protocol or of ICH GCP.

Within 1 year after trial termination the Sponsor will submit a summary of the CTR covering all relevant results of the trial to the Competent Authority and to the Independent Ethics Committee.

The Boehringer Ingelheim transparency and publication policy can be found on the following web page: trials.boehringer-ingelheim.com. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract. As a general rule, no trial results should be published prior to archiving of the CTR.

The terms and conditions of the insurance coverage are made available to the investigator and the subjects, and are stored in the ISF.

#### 8.1 TRIAL APPROVAL, SUBJECT INFORMATION, INFORMED CONSENT

This trial will be initiated only after all required legal documentation has been reviewed and approved by the respective Institutional Review Board (IRB / Independent Ethics Committee (IEC and competent authority (CA) according to national and international regulations. The same applies for the implementation of changes introduced by amendments. Prior to a subject's participation in the trial, written informed consent must be obtained from each subject (or the subject's legally accepted representative) according to ICH-GCP and to the regulatory and legal requirements of the participating country. Each signature must be personally dated by each signatory and the informed consent and any additional subject-information form retained by the investigator as part of the trial records. A signed copy of the informed consent and any additional subject information must be given to each subject or the subject's legally accepted representative.

The subject must be given sufficient time to consider participation in the trial. The investigator or delegate obtains written consent of the subject's own free will with the informed consent form after confirming that the subject understands the contents. The investigator or delegate must sign (or place a seal on) and date the informed consent form. If a trial collaborator has given a supplementary explanation, the trial collaborator also signs (or places a seal on) and dates the informed consent.


Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Re-consenting may become necessary when new relevant information becomes available and should be conducted according to the sponsor's instructions.

The consent and re-consenting process should be properly documented in the source documentation.

#### 8.2 DATA QUALITY ASSURANCE

A risk-based approach is used for trial quality management. It is initiated by the assessment of critical data and processes for trial subject protection and reliability of the results as well as identification and assessment of associated risks. An Integrated Quality and Risk Management Plan documents the rationale and strategies for risk management during trial conduct including monitoring approaches, vendor management and other processes focusing on areas of greatest risk.

Continuous risk review and assessment may lead to adjustments in trial conduct, trial design or monitoring approaches.

A quality assurance audit/inspection of this trial may be conducted by the sponsor, sponsor's designees, or by IRB / IEC or by regulatory authorities. The quality assurance auditor will have access to all medical records, the investigator's trial-related files and correspondence, and the informed consent documentation of this clinical trial..

#### 8.3 RECORDS

CRFs for individual subjects will be provided by the sponsor. For drug accountability, refer to Section 4.1.8.

#### **8.3.1** Source documents

In accordance with regulatory requirements, the investigator should prepare and maintain adequate and accurate source documents and trial records for each trial subject that include all observations and other data pertinent to the investigation. Source data as well as reported data should follow the 'ALCOA principles' and be <u>attributable</u>, <u>legible</u>, <u>contemporaneous</u>, <u>original</u>, and <u>accurate</u>. Changes to the data should be traceable (audit trail).

Data reported on the CRF must be consistent with the source data or the discrepancies must be explained.

Before providing any copy of subjects' source documents to the sponsor, the investigator must ensure that all subject identifiers (e.g., subject's name, initials, address, phone number, and social security number) have properly been removed or redacted to ensure subject confidentiality.

If the subject is not compliant with the protocol, any corrective action (e.g. re-training) must be documented in the subject file.

For the CRF, data must be derived from source documents, for example:

• Subject identification: sex, year of birth (in accordance with local laws and regulations)

c32737758-02

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

- Subject participation in the trial (substance, trial number, subject number, date subject was informed)
- Dates of subject's visits, including dispensing of trial medication
- Medical history (including trial indication and concomitant diseases, if applicable)
- Medication history
- AEs and outcome events (onset date [mandatory], and end date [if available])
- SAEs (onset date [mandatory], and end date [if available])
- Concomitant therapy (start date, changes)
- Originals or copies of laboratory results and other imaging or testing results, with proper documented medical evaluation (in validated electronic format, if available)
- ECG results (original or copies of printouts)
- Completion of subject's participation in the trial (end date; in case of premature discontinuation, document the reason for it, if known)
- Prior to allocation of a subject to a treatment into a clinical trial, there must be documented evidence in the source data (e.g. medical records) that the trial participant meets all inclusion criteria and does not meet any exclusion criteria. The absence of records (either medical records, verbal documented feedback of the subject or testing conducted specific for a protocol) to support inclusion/exclusion criteria does not make the subject eligible for the clinical trial.

#### 8.3.2 Direct access to source data and documents

The investigator /institution will allow site trial-related monitoring, audits, IRB / IEC review and regulatory inspections. Direct access must be provided to the CRF and all source documents/data, including progress notes, copies of laboratory and medical test results, which must be available at all times for review by the Clinical Research Associate, auditor and regulatory inspector (e.g. FDA). They may review all CRFs and informed consents. The accuracy of the data will be verified by direct comparison with the source documents described in Section 8.3.1. The sponsor will also monitor compliance with the protocol and GCP.

#### 8.3.3 Storage period of records

#### Trial site:

The trial site(s) must retain the source and essential documents (including ISF) according to contract or the local requirements valid at the time of the end of the trial (whatever is longer).

#### Sponsor:

The sponsor must retain the essential documents according to the sponsor's SOPs.

#### 8.4 EXPEDITED REPORTING OF ADVERSE EVENTS

BI is responsible to fulfil their legal and regulatory reporting obligation in accordance with regulatory requirements.

c32737758-02 Trial Protocol


Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 8.5 STATEMENT OF CONFIDENTIALITY AND SUBJECT PRIVACY

Individual subject data obtained as a result of this trial is considered confidential and disclosure to third parties is prohibited with the exceptions noted in Section 8.7.

Data protection and data security measures are implemented for the collection, storage and processing of patient data in accordance with the principles 6 and 12 of the WHO GCP handbook.

Personalised treatment data may be given to the subject's personal physician or to other appropriate medical personnel responsible for the subject's welfare. Data generated at the site as a result of the trial need to be available for inspection on request by the participating physicians, the sponsor's representatives, by the IRB / IEC and the regulatory authorities.

# 8.5.1 Collection, storage and future use of biological samples and corresponding data

Measures are in place to comply with the applicable rules for the collection, storage and future use of biological samples and clinical data, in particular

- Sample and data usage has to be in accordance with the informed consent
- The BI-internal or external facilities storing biological samples from clinical trial participants are qualified for the storage of biological samples collected in clinical trials.
- An appropriate sample and data management system, incl. audit trail for clinical data and samples to identify and destroy such samples according to ICF is in place
- A fit for the purpose documentation (e.g. biomarker proposal, analysis plan and report) ensures compliant usage
- A fit for purpose approach will be used for assay/equipment validation depending on the intended use of the data

Samples and/or data may be transferred to third parties and other countries as specified in the ICF.

#### 8.6 TRIAL MILESTONES

The **start of the trial** is defined as the date of the enrolment of the first subject in the trial.

The **end of the trial** ('Last Subject Completed') is defined as the 'date of the last visit of the last subject in whole trial'.

Early termination of the trial is defined as the premature termination of the trial for any reason before the end of the trial as specified in this protocol.

**Temporary halt of the trial** is defined as any unplanned interruption of the trial by the sponsor with the intention to resume it.

**Suspension of the trial** is defined as an interruption of the trial based on a Health Authority request.

The EC/competent authority in each participating EU member state will be notified about the trial milestones according to the laws of each member state.


Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

A final report of the clinical trial data will be written only after all subjects have completed the trial in all countries (EU or non-EU), so that all data can be incorporated and considered in the report.

The sponsor will submit to the EU database a summary of the final trial results within one year from the end of a clinical trial as a whole, regardless of the country of the last patient (EU or non-EU).

#### 8.7 ADMINISTRATIVE STRUCTURE OF THE TRIAL

The trial is sponsored by Boehringer Ingelheim.

The trial will be conducted at under the supervision of the Principal Investigator. Tasks and responsibilities are defined in a contract. Relevant documentation on the participating (Principal) Investigators (e.g. their curricula vitae) will be filed in the ISF.

BI has appointed a Clinical Trial Leader, responsible for coordinating all required trial activities, in order to

- Manage the trial in accordance with applicable regulations and internal SOPs
- Direct the clinical trial team in the preparation, conduct, and reporting of the trial
- ensure appropriate training and information of local clinical monitors (CML), Clinical Research Associates, and investigators of participating trial sites

The trial medication will be provided by the (BI 706321) or will be obtained by the clinical trial site from public pharmacy (itraconazole).

Safety laboratory tests will be performed by the local laboratory of the trial site

Analyses of BI 706321 concentrations in plasma will be performed at

On-site monitoring will be performed by BI or a contract research organisation appointed by BI.

Data management and statistical evaluation will be done by BI or a contract research organisation according to BI SOPs.

Tasks and functions assigned in order to organise, manage, and evaluate the trial are defined according to BI SOPs. A list of responsible persons and relevant local information can be found in the ISF.

c32737758-02 Trial Protocol 

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 9. REFERENCES

#### 9.1 PUBLISHED REFERENCES

| P07-13746 | Heeswijk RPG van, Bourbeau M, Campbell P, Seguin I, Chauhan BM, Foster BC, Cameron DW. Time-dependent interaction between lopinavir/ritonavir and fexofenadine. J Clin Pharmacol 46, 758-767 (2006). |
|---|---|
| P15-06298 | Ministry of Health, Labour and Welfare. Drug interaction guideline for drug development and labeling recommendations (draft).<br>http://www.solvobiotech.com/documents/Japanese_DDI_guideline_(draft) _2014Jan.pdf (access date: 22 June 2015); Ministry of Health, Labour and Welfare; 2014. |
| P15-06991 | European Medicines Agency (EMA). Committee for Human Medicinal Products (CHMP): guideline on the investigation of drug interactions (21 June 2012, CPMP/EWP/560/95/rev. 1 corr. 2). http://www.ema.europa.eu/docs/en_GB/document_library/Scientific_guideline/2012/07/WC500129606.pdf (access date: 8 July 2015); London: European Medicines Agency (EMA); 2012. |
| R01-0516 | Olkkola KT, Backman JT, Neuvonen PJ. Midazolam should be avoided in patients receiving the systemic antimycotics ketoconazole or itraconazole. Clin Pharmacol Ther 1994. 55(5):481-485. |
| R08-1652 | Kharasch ED, Bedynek PS, Walker A, Whittington D, Hoffer C. Mechanism of ritonavir changes in methadone pharmacokinetics and pharmacodynamics: II. Ritonavir effects on CYP3A and P-glycoprotein activities. Clinical Pharmacology and Therapeutics, advance online publication 9 July 2008, doi:10.1038/clpt.2008.102 Clin Pharmacol Ther 2008. |
| R10-1102 | Templeton IE, Thummel KE, Kharasch ED, Kunze KL, Hoffer C, Nelson WL, Isoherranen N. Contribution of itraconazole metabolites to inhibition of CYP3A4 in vivo. Clin Pharmacol Ther 2008; 83(1):77-85. |
| R11-5230 | Julious SA. Sample sizes for clinical trials. Boca Raton: Taylor & Francis Group; 2010. |
| R12-1392 | Levey AS, Stevens LA, Schmid CH, Zhang Y, Castro AF, Feldman HI, Kusek JW, Eggers P, Lente F van, Greene T, Coresh J, Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI). A new equation to estimate glomerular filtration rate. Ann Intern Med 2009;150(9):604-612. |
| R15-3252 | Jalava KM, Partanen J, Neuvonen PJ. Itraconazole decreases renal clearance of digoxin. Ther Drug Monit 1997. 19(6):609-613. |

c32737758-02 Trial Protocol 

| Proprietary confidentia | al information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies |
|---|---|
| R17-3742 | Barone JA, Moskovitz BL, Guarnieri J, Hassell AE, Colaizzi JL, Bierman RH, et al. Food interaction and steady-state pharmacokinetics of itraconazole oral solution in healthy volunteers (2017). Pharmacotherapy 1998; 18(2); 295-301. |
| R17-3743 | Willems L, Geest R van der, Beule K de. Itraconazole oral solution and intravenous formulations: a review of pharmacokinetics and pharmacodynamics. J Clin Pharm Ther 2001; 26:159-169. |
| R17-3744 | Liu L, Bello A, Dresser MJ, Heald D, Komjathy SF, O'Mara E, et al. Best practices for the use of itraconazole as a replacement for ketoconazole in drug-drug interaction studies. J Clin Pharmacol 2016. 56(2):143-151. |
| R18-0241 | Guidance for industry: clinical drug interaction studies - study design, data analysis, and clinical implications (draft guidance, this guidance document is being distributed for comment purposes only) (October 2017, clinical pharmacology). https://www.fda.gov/downloads/drugs/guidances/ucm292362.pdf (access date: 19 January 2018); Silver Spring: U.S. Department of Health and Human Services, Food and Drug Administration, Center for Drug Evaluation and Research (CDER) 2017. |
| R18-2643 | Sporanox 10 mg/ml oral solution (Janssen-Cilag) (summary of product characteristics, updated 01-Mar-2018). https://www.medicines.org.uk/emc/product/1522/smpc/print (access date: 14 August 2018); 2018. |

| R20-2709 | Sempera Liquid 10 mg/ml, Loesung zum Einnehmen (Janssen-Cilag) (Fachinformation, Stand der Information: May 2020). 2020. |
|---|---|
| R94-1529 | Chow SC, Liu JP, editors. Design and analysis of bioavailability and bioequivalence studies. New York: Marcel Dekker Inc., 1992. |

# 9.2 UNPUBLISHED REFERENCES

| 001-MCS-36-472 | Standards and processes for analyses performed within Clinical Pharmacokinetics/Pharmacodynamics. Current version |
|---|---|
| c02336088 | Relative bioavailability of a single oral dose of BI 691751 when administered alone or in combination with multiple oral doses of itraconazole in healthy male subjects (an openlabel, randomised, two-period, two-sequence crossover study). Clinical Trial Report. 1334.10. 09 January 2015. |
| c03355329 | Relative bioavailability of a single oral dose of BI 425809 when administered alone or in combination with multiple oral doses of itraconazole in healthy male subjects (an openlabel, two-period, fixed-sequence trial). Clinical Trial Report. 1346.10. 03 December 2015. |

Boehringer Ingelheim BI Trial No.: 1425-0010 01 Feb 2021

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

c08928447

Effect of multiple doses of itraconazole on the pharmacokinetics of a single oral dose of BI 1026706 in healthy male subjects (an open-label, randomised, two-period, two-sequence crossover study). Clinical Trial Report. 1320.20. 29 September 2016.

**Boehringer Ingelheim** BI Trial No.: 1425-0010

01 Feb 2021

**Trial Protocol** 

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### **APPENDICES 10.**

Not applicable.

c32737758-02


c32737758-02 Trial Protocol 

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 11. DESCRIPTION OF GLOBAL AMENDMENT(S)

#### 11.1 GLOBAL AMENDMENT 1

| Date of amendment | 01 February 2021 |
|---|---|
| EudraCT number | 2020-004388-22 |
| BI Trial number | 1425-0010 |
| BI Investigational Medicinal Product | BI 706321 |
| Title of protocol | Effect of itraconazole on the pharmacokinetics of a single oral dose of BI 706321 in healthy male subjects (an open-label, two-period fixed sequence design study) |
| To be implemented only after approval of the IRB / IEC / Competent Authorities To be implemented immediately in order to eliminate hazard – IRB / IEC / | |
| | Competent Authority to be notified of change with request for approval Can be implemented without IRB / IEC / Competent Authority approval as |
| changes involve logistical or ac | <u> </u> |
| onwiges my orver registrous or wi | warning war to dispect to only |
| Section to be changed | 5.3.2.1 |
| Description of change | Changed handling of PK blood samples taken for analysis of BI 706321 (allowed time period between sample withdrawal and freezing shortened; interim storage of blood samples on ice instead of at room temperature) |
| Rationale for change | Unknown stability data in case of further use of samples (e.g. metabolite determination) |



#### APPROVAL / SIGNATURE PAGE

Document Number: c32737758 Technical Version Number: 2.0

**Document Name:** clinical-trial-protocol-version-02

**Title:** Effect of itraconazole on the pharmacokinetics of a single oral dose of BI 706321 in healthy male subjects (an open-label, two-period fixed sequence design study)

# **Signatures (obtained electronically)**

| Meaning of Signature | Signed by | Date Signed |
|---|---|---|
| Author-Clinical Trial Leader | | 01 Feb 2021 17:19 CET |
| Approval-Team Member Medicine | | 01 Feb 2021 17:36 CET |
| Author-Trial Statistician | | 02 Feb 2021 09:22 CET |
| Verification-Paper Signature<br>Completion | | 02 Feb 2021 13:46 CET |
| Approval-Clinical Pharmacokinetics | | 04 Feb 2021 20:15 CET |
| Approval-Therapeutic Area | | 08 Feb 2021 17:49 CET |

Boehringer IngelheimPage 2 of 2Document Number: c32737758Technical Version Number: 2.0

(Continued) Signatures (obtained electronically)

| Meaning of Signature | Signed by | Date Signed |
|----------------------|-----------|-------------|
|----------------------|-----------|-------------|